

| Official Title: | PT4A (Peers and Technology for Adherence, Access, Accountability, and Analytics) - A Qualitative Study |
|---|---|
| NCT Number: | NCT05051124 |
| Study Number: | 20-01579 |
| Document Type: | Study Protocol and Statistical Analysis Plan |
| Date of the Document: | • December 23, 2022 |

# PEERS AND TECHNOLOGY FOR ADHERENCE, ACCESS, ACCOUNT-ABILITY, AND ANALYTICS (PT4A)

### <u>PI</u>

Dr. Rajesh Vedanthan, MD, MPH

### CO-Is

Dr. Benson Njuguna, B. Pharm, MPPM

Dr. Sonak Pastakia, PharmD, MPH, BCPS

Dr. Tina Tran, PharmD

Dr. Jeremiah Laktabai, MD

Dr. Juddy Wachira, PhD

Dr. Ann Mwangi, PhD

Dr. Imran Manji, B. Pharm, MPH

Dr. Antoinette Schoenthaler, EdD

Dr. Andrea Troxel, ScD

Dr. Becky Genberg, PhD

Dr. Dustin Duncan, ScD

### CONTENTS

### **CONTENTS**

| STATEMENT OF COMPLIANCE | 2 |
|---|---|
| PROTOCOL SYNOPSIS | 4 |
| SIGNIFICANCE | 7 |
| INNOVATION | 9 |
| APPROACH | 9 |
| Preliminary Data | 10 |
| International Advisory Committee | 11 |
| Overall Implementation Research Framework | 12 |
| Aim 1: Identify micro- and macro-level contextual factors that might influence the implementation of the PT4A strategySub Aim 2.1: Evaluate The Intervention For Accel And Appropriateness | |
| Rigor and Reproducibility | 19 |
| Assessment of Potential Risks and Benefits | 20 |
| Milestones | 25 |
| Table 4: PT4A Milestones | 27 |
| Timeline | 27 |
| REFERENCES | 28 |
| APPENDIX A | 37 |
| PT4A AIM 2 STUDY PROTOCOL | 37 |
| APPENDIX B | 47 |
| STUDY INTERVIEW QUESTIONNAIRES | 47 |
| APPENDIX C | 59 |

### STATEMENT OF COMPLIANCE

The trial will be carried out in accordance with International Council on Harmonization Good Clinical Practice (ICH GCP) and the following:

• United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 312, and/or 21 CFR Part 812).

National Institutes of Health (NIH)-funded investigators and study site staff who are responsible for the conduct, management, or oversight of the study have completed Human Subjects Protection and ICH GCP Training.

### PROTOCOL SYNOPSIS

| Title: | Peers and Technology for Adherence, Access, Accountability, |
|---|---|
| O (N) | and Analytics (PT4A) – A Qualitative Study |
| Grant Number: | 1R56HL150036 |
| Study Description: | The overall objective of this project is to utilize the PRECEDE-PROCEED framework to conduct transdisciplinary, translational implementation research focused on improving medication adherence for hypertension control. The central hypothesis is that peer delivery of medications integrated with HIT (PT4A) will be effective in improving hypertension medication adherence, contributing to improved blood pressure among patients with uncontrolled hypertension in western Kenya. This application will focus on the critical formative components of the overall implementation research objective, and we propose the following specific aims: Aim 1 will identify micro- and macro-level contextual factors that might influence the implementation of the PT4A strategy (individual, family, clinician, health system, and environment), using qualitative methods. Aim 2: We will then use a humancentered design approach to refine the PT4A intervention using the findings from Aim 1. Sub-Aim 2.1 will evaluate the intervention for acceptability and appropriateness by use of a survey tool with patients, peers, and clinical staff. In Sub-Aim 2.2, we will then conduct a pilot of the intervention and conduct a survey questionnaire with patients, peers, and clinical staff to evaluate feasibility. We will evaluate impact on systolic blood pressure, medication adherence, and fidelity of implementation. We will also create a retrospective comparator (control) group of CDM patients, through querying AMRS, matched by sex, age, location and initial blood pressure level. We will then use their recorded blood pressure over a comparable period of upto 1 year and to allow for comparison to the blood pressure changes observed in the patients enrolled in the PT4A program to help understand the magnitude and variance of the intervention effects. |
| Objectives*: | The overall objective of this proposal is to utilize transdisciplinary, translational implementation research, guided by the PRECEDE-PROCEED framework, to address the challenge of hypertension medication non-adherence in low-resource settings. |
| Endpoints*: | The <u>primary adherence outcome</u> is the pill count adherence ratio, which is the proportion of prescribed doses taken over a 1-month time period, assessed at the end of the pilot. The <u>primary implementation outcome</u> is fidelity, measured as quantity and quality of intervention delivery as intended, comprised of three components: confirmed medication delivery documented by patient e-signature, peer completion of the HIT form, and quality of data entry into the HIT form. |

| | T |
|---|---|
| Study Population: | Approximately 146 individuals will participate in this study. The number is approximate because for focus group discussions, the number of participants can range from 6-10. Aim 1: • Focus group discussions (approximately 96 participants): Participants will be patients with hypertension who are currently enrolled in the AMPATH CDM program, and at least 18 years of age from the counties of Bungoma, Trans Nzoia, and Uasin Gishu in Western Kenya. Clinical staff in the AMPATH CDM program and community leaders from the counties will also participate. (12 total FGDs, 6-10 participants each) • Key informant interviews (4 participants): Participants will be County Executive Committee representatives for health from the three Counties included in the study and the Ministry of Health head for non-communicable diseases (NCDs). |
| | Aim 2: • Human Centered Design Team (20 participants): Participants will be individuals representing the following stakeholder groups: research team members, clinicians, pharmacists, peers, patients with hypertension, representatives from the informatics team, and other relevant staff members involved in hypertension care Aim 2.1: |
| | <ul> <li>Use of Survey tools adapted from acceptability and appropriateness measures (39 participants):</li> <li>Participants will be patients (as described above), peer navigators, and clinical staff (as described above).</li> <li>Aim 2.2:</li> <li>Pilot (up to 100 participants): Participants will be patients who are currently enrolled in the AMPATH CDM program, and at least 18 years of age from the counties of Bungoma, Trans Nzoia, and Uasin Gishu in</li> </ul> |
| | <ul> <li>Western Kenya.</li> <li>Retrospective comparator group: AMRS records of up to<br/>100 patients who will serve as a control group matched<br/>by sex, age, location and initial blood pressure level</li> </ul> |
| Phase* or Stage: | N/A |
| Description of | AMPATH catchment area in three counties of western Kenya: |
| Sites/Facilities Enrolling Participants: | Bungoma, Trans Nzoia, and Uasin Gishu. |

| Description of Study | Peer delivery of medications: We will adopt a novel approach of |
|---|---|
| Intervention/Experimental | extending beyond the use of peer support in the clinical setting |
| Manipulation: | |
| | extending beyond the use of peer support in the clinical setting and implement door-to-door peer delivery of medications within atients' communities lealth Information Technology (HIT) Platform: To support peer elivery, we will use a HIT platform that performs 4 core unctions: 1) tailored counseling strategies through decision upport; 2) teleconsultation support for clinician-peer-patient ateractions; 3) tracking medication refills to enhance occountability of the peer delivery process; and 4) analytics to approve medication supply chain by generating patient-level |
| | and implement door-to-door peer delivery of medications within atients' communities <u>ealth Information Technology (HIT) Platform:</u> To support peer delivery, we will use a HIT platform that performs 4 core notions: 1) tailored counseling strategies through decision upport; 2) teleconsultation support for clinician-peer-patient teractions; 3) tracking medication refills to enhance ecountability of the peer delivery process; and 4) analytics to approve medication supply chain by generating patient-level |
| | delivery, we will use a HIT platform that performs 4 core |
| | functions: 1) tailored counseling strategies through decision |
| | pport; 2) teleconsultation support for clinician-peer-patient eractions; 3) tracking medication refills to enhance |
| | eractions; 3) tracking medication refills to enhance |
| | ccountability of the peer delivery process; and 4) analytics to |
| | improve medication supply chain by generating patient-level |
| | drug consumption data. This is an innovative use of HIT to |
| | accomplish these functions to support medication adherence. |
| Study Duration*: | Up to 1 year |
| Participant Duration: | Up to 1 year |

### A. SIGNIFICANCE

<u>Hypertension – Global Burden and Unmet Needs.</u> Elevated blood pressure (BP) is the leading risk factor of death globally. The global burden of hypertension is increasing, disproportionately so in low- and middle-income countries (LMICs). While BP control reduces cardiovascular disease (CVD) and death, treatment and control rates remain suboptimal both in the U.S. and LMICs. The economic burden of hypertension is staggering, in terms of both direct health costs and indirect impact on employment and productivity. Despite many evidence-based interventions to manage hypertension, substantial implementation gaps persist.

Medication Adherence. Adherence is defined as "the process by which patients take their medications as prescribed," and is often divided into three phases: initiation, implementation, and persistence. Adherence to hypertension medication reduces congestive heart failure, 19 CVD risk, 20 CVD events, 21,22 and mortality. 21-24 Despite increased medication costs, adherence can lead to net decrease in both health care utilization and cost in hypertensive patients. Siven the clinical and economic benefits of adherence, improvements in hypertension medication adherence will improve BP control and reduce CVD risk and mortality. However, in low-resource settings worldwide, nearly 60% of hypertension patients report non-adherence to antihypertensive medications—both suboptimal implementation (i.e. day-to-day medication-taking behavior) and non-persistence (i.e. premature discontinuation), leading to poor BP control and increased hospitalization and mortality. 27-33

Multi-Level Barriers Impacting Adherence. Barriers to adherence to hypertension medications are complex and multi-level. 32,34-37 At the macro-level (e.g. health systems and communities), challenges include reduced medication availability, 38 low affordability, 38 inadequate insurance coverage, 32 transportation, 39,40 and distance to health facilities. 41,42 At the micro-level (e.g. individual patients and providers), barriers include provider training, 43 poor patient-provider relationships, 44-46 patient missing doses, 40 real and perceived adverse effects, 47 and psychological factors. 40,48 Therefore, there is a need to develop and evaluate rigorous implementation strategies that address the multi-level barriers impacting medication adherence.

<u>Peer Delivery of Medications.</u> Peers are lay individuals with shared disease experience who provide practical, social, emotional, and motivational assistance to patients. <sup>49</sup> Peer support can improve chronic disease medication adherence; however, most studies have occurred in clinical settings. <sup>50-52</sup> <u>To date, door-to-door peer delivery of hypertension medications to patients in order to improve adherence has not been evaluated.</u>

<u>Health Information Technology (HIT).</u> The use of HIT, such as electronic medical record systems, mobile health (mHealth) approaches, and electronic prescribing, can enhance medication adherence. In LMICs, HIT has demonstrated beneficial impact on clinical care processes for chronic diseases, and can enhance peer support networks for non-communicable disease (NCD) care. However, it is not well known if HIT, combined with peer delivery, can enhance adherence to antihypertensive medications and improve BP control. S8,59

<u>Rigor of Prior Research.</u> As described above, a large evidence base has clearly documented that medication adherence is associated with improved BP and CVD outcomes. However, micro- and macro-level barriers to hypertension medication adherence lead to suboptimal BP control and adverse CVD outcomes. While peer support and HIT have separately shown promise with respect to improving medication adherence, there remain gaps in the literature that will be addressed by our proposed project to combine peer delivery and HIT to address multiple barriers, thereby improving hypertension medication adherence, ultimately contributing to improved BP among patients with uncontrolled hypertension in western Kenya.

Relevance to the U.S. The burden of hypertension in the U.S. is substantial, 60 and the challenges for population subgroups (health facility access, transportation, and opportunity cost of lost work) are similar to those in Kenya. 61 Despite efforts to improve adherence, gaps remain leading to morbidity, mortality, and costs. 62 Hence, we aim to produce generalizable knowledge relevant to the U.S. In fact, our team and colleagues have previously translated research learnings from Kenya into impactful interventions for U.S. communities. 63-65

Implementation Science Training and Capacity Building. Capacity building has been a longstanding priority for our team and is fundamental to this project. 66-73 We are therefore purposely involving a relatively junior Kenyan sub-award investigator with more experienced U.S.-based Multiple Principal Investigators. In addition to this experiential learning, we will leverage didactic training activities, as we have previously done. This human resource investment will ensure future implementation research related to hypertension and other NCDs.

### **B. INNOVATION**

<u>Human-Centered Implementation Research.</u> Human-centered design (HCD) is a creative approach to problem-solving, a process whereby stakeholders are engaged in all phases: inspiration (identify the challenge), ideation (design, test and refine solutions) and implementation (maximize impact).<sup>76,77</sup> Our team has previously utilized HCD in the context of NCD care and prevention, and we have previously proposed an approach termed "human-centered implementation research".<sup>78-81</sup> Using this approach is pioneering and could provide a model for co-creation and participatory design that could be relevant worldwide.

<u>Peer Delivery of Medications.</u> We will adopt a novel approach of extending beyond the use of peer support in the clinical setting and implement door-to-door peer delivery of medications within patients' communities.

<u>Health Information Technology (HIT) Platform.</u> To support peer delivery, we will use a HIT platform that performs 4 core functions: 1) <u>tailored counseling strategies</u> through decision support; 2) <u>teleconsultation</u> support for clinician-peer-patient interactions; 3) tracking medication refills to enhance <u>accountability of the peer delivery process</u>; and 4) <u>analytics to improve medication supply chain</u> by generating patient-level drug consumption data. This is an innovative use of HIT to accomplish these functions to support medication adherence.

### C. APPROACH

<u>Setting.</u> The proposed study will take place in western Kenya at the Academic Model Providing Access to Healthcare (AMPATH) program, an academic partnership between Moi University College of Health Sciences (MUCHS), Moi Teaching and Referral Hospital (MTRH), and a consortium of North American universities. AMPATH has established an HIV care program that has enrolled over 200,000 patients in a catchment population of 4 million. AMPATH was designated as a Center of Excellence for Cardiovascular and Pulmonary Disease Research by the NHLBI. At the same time, AMPATH also established a Chronic Disease Management (CDM) Program in collaboration with the Ministry of Health (MOH). We have a Memorandum of Understanding with the Kenya MOH to provide care for NCDs and to develop and evaluate innovative approaches to NCD management including hypertension.

The CDM Program has enrolled over 40,000 patients with hypertension. Our team has conducted several NIH-funded implementation research studies targeting various elements of the NCD care delivery system: nurse management of hypertension (K01TW009218), linkage/retention to hypertension care (U01HL114200), group medical visits and microfinance for NCDs (R01HL125487), and strengthening referral networks for hypertension (U01HL138636). In addition, we have implemented a network of revolving fund pharmacies (RFPs) to ensure a reliable supply of medicines for hypertension and other NCDs across all levels of the health system, including 60 health facilities where availability of medications for hypertension is now 95-99%. 35,86-88

AMPATH has used the AMPATH Medical Records System (AMRS), a customized version of OpenMRS, since 2005. 89 In 2016, AMPATH developed a software program called "Point-of-Care" (AMRS-POC), which we started using in CDM clinics for hypertension management in 2017. We have developed software modules for the following clinical functions: 1) historical patient data review (patient dashboard); 2) real-time clinical data entry (customized interactive forms with skip logic); 3) decision support tailored to the type and training of clinician (e.g. when to escalate hypertension therapy); 4) health facility management (scheduling, follow-up of patients missing clinic visits, generating administrative reports); and 5) data visualization (quality indicators). AMPATH has invested in a Wi-Fi network and solar power system to ensure network access and server connectivity for each health facility. Our current system is being

implemented in over 30 health facilities serving a patient population of nearly 100,000 patients, and has been used for more than 1 million clinical encounters. We have developed and implemented a HIT-based home glucose monitoring program that has led to significant improvements in glycemic control. We have also implemented real-time interactive HIT for oncology, enabling specialists at the referral hospital to co-manage patients with clinicians from remote health facilities. Finally, we are developing a personal health record platform to support asynchronous telemedicine. The proposed HIT component of this study builds upon this established infrastructure.

### **Preliminary Data.**

<u>Suboptimal Medication Adherence</u>. Adherence to hypertension medications is suboptimal in western Kenya, and there remain gaps to improve patient-level access and medication refill rates. Preliminary analysis of data from participants in the BIGPIC trial (R01HL125487) indicates that <u>nearly 50% of patients</u> with hypertension and/or diabetes reported suboptimal adherence, similar to other countries in Africa.<sup>37</sup> Due to limited cash supply, patients often choose to fill only a part of their prescription on the day of the clinic visit, and are expected to return for refills. AMPATH pharmacy data indicate that as the prescription duration increases, fewer patients fill the prescription for the entire period: 43% filled their 60-day prescription, and only 21% filled their 90-day prescription. The remaining patients required a return visit to refill their prescriptions. However, missed refills are frequent; in fact, 62% of hypertensive patients in this region reported having missed or skipped a refill, while 64% reported having run out of medication before the next refill date. Pharmacy program data confirm this self-report; a recent audit indicated that only 24% of individuals who were due to return to clinic for a prescription refill actually did

Figure 1. Study sites in western Kenya



SO.

Impact of Adherence on BP. Suboptimal adherence in our catchment is associated with worse BP outcomes: individuals reporting having missed doses of medications had an average systolic BP (SBP) of 157 mmHg compared to 134 mmHg among those with perfect adherence. Those who had run out of medications and missed refills also had higher SBP levels (unpublished data).

<u>Factors Impacting Adherence</u>. For hypertension patients in Kenya, unaffordability of care, low availability of providers, poor access to health facilities, and inadequate social support are all barriers to hypertension care and medication adherence.<sup>42,91</sup> Cost of transport and distance to

the health facility have also been reported as significant barriers. Preliminary analysis of BIGPIC trial data indicates that time taken to reach the health facility is significantly associated with a missed prescription;<sup>79</sup> round-trip estimates average approximately 90-120 minutes. In addition, patients spend nearly two hours at the health facility when attending a hypertension clinic, or even just for a medication refill. We have previously reported that the clinician-patient encounter averages less than 10 minutes,<sup>92</sup> indicating long wait times and therefore time lost from work. To supplement the substantive preliminary data summarized above, we propose to conduct a more thorough assessment of the various factors that might impact successful implementation of the PT4A strategy.

Results from Peer and HIT Involvement in Care Delivery. We have successfully used peers in the AMPATH program to provide adherence counseling and psychosocial support for patients with HIV.<sup>93,94</sup> We have also delivered portable group-based NCD care, peer support, and medications in remote, patient-centered locations for several years, with improvements in retention in PT4A Protocol 1.4 23<sup>rd</sup> November, 2022

| Table 1: Investigator expertise in proposed | work |
|---|---|
| <u>Domain</u> | <u>Investigators</u> |
| Hypertension management in LMICs | Vedanthan, Pastakia, Njuguna, Tran, Laktabai, Manji |
| Systems improvement in NCD care | Vedanthan, Pastakia, Njuguna, Tran, Laktabai, Manji |
| NCD-related implementation science | Vedanthan, Pastakia, Njuguna, Njuguna, Genberg |
| Peer-based care for hypertension | Vedanthan, Pastakia, Njuguna, Tran |
| Health IT for NCD care | Vedanthan, Pastakia, Njuguna, Dick |
| Expanding access to medications | Vedanthan, Pastakia, Njuguna, Tran, Manji |
| Medication adherence research | Schoenthaler, Genberg |
| Qualitative research | Schoenthaler, Wachira, Genberg |
| Epidemiology | Vedanthan, Genberg |
| Spatial analysis | Duncan |
| Biostatistics and transportability analysis | Troxel, Mwangi |
| Cost effectiveness and decision analysis | Finkelstein |

care, BP, and A1c.<sup>79,95,96</sup> Our program of peer delivery of HIV medications, begun over one year ago, has grown by nearly 20%, with 97% of medications delivered on time. We also have implemented a pilot program of peer delivery of medications for hypertension and diabetes, with improvement in adherence and a nearly 6-mmHg reduction in SBP. We have also shown that HIT strategies can integrate and coordinate care across the

health system for HIV, diabetes, and hypertension.85,97-100

Summary of Preliminary Data and Remaining Gaps. As described above, the current proposal is an extension of established work, building upon a solid foundation of several years and iterations of peer- and HIT-based strategies. However, there remain implementation gaps, as well as gaps in the rigor of prior research, to be addressed. We hypothesize that our proposed strategy, peers and technology for adherence, access, accountability, and analytics (PT4A), will help to address some of the remaining gaps we have identified in our prior research. As an initial step, further formative research is required prior to full-scale implementation and evaluation of this strategy to improve medication adherence and blood pressure. We will conduct this project in the AMPATH catchment area in three counties of western Kenya: Bungoma, Trans Nzoia, and Uasin Gishu (Figure 1).

Study Team. Our proposal builds upon longstanding institutional partnerships that comprise the AMPATH Consortium, which have laid the groundwork for clinical care and research in CVD. 67,82,84,85,101-103 Both Dr. Vedanthan (contact PI) and Dr. Pastakia (MPI) have successfully collaborated for several years with each other and with investigators from MUCHS and MTRH, as well as members of the current study team, to establish robust structures for chronic disease research and clinical care in western Kenya. 67,68,79,85,91,99,104-109 Each collaborator adds specific value to this proposal (Table 1). Critically, we have secured strong high-level political support from the Head of the Division of NCDs at the MOH. In addition, the AMPATH Executive Director of Care is supportive of this application. The head of the AMPATH Population Health Program, Dr. Laktabai, as well as the head of the AMPATH RFP program, Imran Manji, are co-investigators. This key program and government leadership support provide a strong foundation that positions us to successfully carry out our proposed research and produce lessons and insights that can have impact worldwide.

<u>International Advisory Committee.</u> Our goal is to make the PT4A strategy relevant for health systems in low-resource settings worldwide. We will therefore create an International Advisory Committee consisting of peers, researchers, clinicians, administrators, and policy makers from around the world. Twice a year, the committee will discuss by teleconference how to tailor the strategy for the Kenyan context as well as in other low-resource settings, and how to adapt, implement, and evaluate the PT4A strategy in other contexts.

<u>Stakeholder Engagement.</u> We will collaborate with key stakeholders throughout the proposed project. At the **conception** stage, we have aligned our proposal to address a key national priority: curbing NCDs while addressing the shortage of human resources for health. We have also already secured input and support for this proposal from the MOH NCD leadership. At the **design** phase, we have engaged key program leaders both informally and formally as

PT4A Protocol 1.4 23<sup>rd</sup> November, 2022

investigators on this proposal, leveraging their experience with NCD care, peer-based care, and NCD medication adherence, thus ensuring our proposed strategy is aligned with program and policy priorities. <sup>83</sup> We will engage patients, communities, clinicians and health program leaders as we **conduct** our qualitative research and human-centered design-based strategy refinement. AMPATH's Community Strategy Initiative routinely engages existing community-based governance structures to gather input and feedback on community-based initiatives. In addition, the AMPATH research program has a long history of engaging and informing community stakeholders of research interventions. <sup>79,108,111-121</sup> finally, we will conduct regular **dissemination** of our program experiences, successes, and challenges to key stakeholders to co-create solutions and promote receptivity for future wider implementation.

<u>Overall Implementation Research Framework.</u> The PRECEDE-PROCEED framework provides a conceptual framework for assessment of an implementation challenge, design of a responsive strategy, and implementation and evaluation of that strategy (Figure 2). 122-124 We



chose to use PRECEDE-PROCEED as our overall implementation research framework because of its participatory nature, multi-pronged assessment of the multi-level factors that affect adherence, and multiple evaluation components. In addition, PRECEDE-PROCEED is appropriate for a hybrid type 2 implementation research trial, 125 where we will have a dual focus to assess effectiveness of the strategy in improving medication adherence and BP, while also evaluating the fidelity of our implementation strategy. We are currently using PRECEDE-PROCEED in another NIH-funded study, 126 while others have successfully used this framework to develop strategies to promote cardiovascular health in low-income populations. 127 Phases 1 and 2 are simultaneous with our baseline contextual assessment (Aim 1). Phase 3 aligns with the HCD

process (Aim 2). Phase 4 aligns with the acceptability, appropriateness, and feasibility testing. Phases 5 to 8 will encompass the subsequent planned R01 grant application. Phase 5 will be the implementation of the cluster randomized trial comparing the PT4A strategy to usual care. Phase 6 will align with our impact and outcome evaluation to determine the overall impact as well as the impact of spatial factors on strategy effect, respectively. The Phase 7 process evaluation will be implemented simultaneous with Phase 5, and Phase 8 is our planned scalability and adaptability evaluation.

Conceptual Model for Adherence Behavior. We will use the capability, opportunity, and motivation model for behavior change (COM-B)<sup>128</sup> as our conceptual model for medication adherence behavior. The COM-B model provides a solid foundation to comprehensively understand the multi-level determinants of adherence, and develop our strategy targeting improved adherence (Table 2). We chose the COM-B model due to its versatility at addressing a variety of behavior change challenges, its applicability in low-resource settings, and its comprehensiveness in recognizing interactions among multiple determinants of the same problem. 106,129-133

We hypothesize that the PT4A strategy will address determinants of hypertension medication adherence at the micro- and macro-levels, leading to changes in patient activation, improvement in adherence, and reduction of BP. Peer-based delivery of medications will reduce both direct costs (e.g. transport) and opportunity costs (e.g. time lost, time off economic activity) associated with acquiring medication refills. Secondly, peer delivery will provide a platform for peer-patient interaction that can be leveraged to provide adherence counseling and psychoso-

| | B constructs, det<br>/I-B Construct | erminants of medication adherence, and propo<br>Determinant of Adherence | psed PT4A intervention components PT4A Intervention Components | port.<br>Through |
|---|---|---|---|---|
| Capability | Physical<br>(Micro) | How and when to take medicines Pill burden | Peer: adherence counseling HIT: decision support and targeted counseling | the inter- |
| | Psychological<br>(Micro) | <ul> <li>Individual knowledge about medicines,<br/>hypertension and adherence necessity</li> <li>Understanding the relationship between<br/>adherence and clinical outcomes</li> </ul> | Peer: adherence counseling<br>HIT: decision support and targeted counseling | action,<br>peers<br>may help |
| Opportunity | Social<br>(Macro) | <ul> <li>Social norms about hypertension and treatment</li> <li>Social support for adherence</li> </ul> | Peer: psychosocial support | address<br>medica- |
| | Physical<br>(Macro) | Time, ease, and cost of transport to acquire refill Availability and price of medications Opportunity cost of acquiring refill | Peer: medication delivery Peer: psychosocial support HIT: teleconsultation HIT: supply chain analytics | tion-re-<br>lated cor<br>cerns |
| Motivation | Reflective<br>(Micro) | <ul> <li>Individual barriers and facilitators of<br/>adherence</li> <li>Individual beliefs about hypertension and<br/>medicines</li> <li>Patient activation in his/her care</li> </ul> | Peer: adherence counseling Peer: psychosocial support Peer: health coaching HIT: decision support and targeted counseling | (e.g. per-<br>ceived<br>and real |
| | A utomatic<br>(Micro) | Habits/Medication routines Emotional response to disease and medicines | Peer: adherence counseling<br>Peer: psychosocial support<br>HIT: decision support and targeted counseling | adverse effects), |

rt. rough e intertion, ers ay help ldress edican-reed conrns g. perived id real lverse fects),

improve patient activation (e.g. coaching patients to raise concerns and questions with clinicians), and provide psychosocial support. HIT will augment peer roles through the decision support system, teleconsultation functionality, and provision of patient-specific adherence summaries for targeted counseling. The HIT platform will also provide enhanced supply chain analytics in order to optimize availability of medications at the rural dispensing facilities.

### Aim 1: Identify micro- and macro-level contextual factors that might influence the implementation of the PT4A strategy.

We will use qualitative research methods to conduct a thorough baseline contextual assessment of barriers and facilitators for implementing PT4A.

Participants: We will conduct focus group discussions (FGDs) of 6-10 participants each among four different groups in each county

: individuals with hypertension (men and women separately), clinical staff, and community members (12 total FGDs). Purposive sampling will be used to select study participants in order to sample a diversity of stakeholders. For individuals with hypertension, diversity of age and distance from the nearest health facility will be targeted. In addition, we will conduct four key informant interviews (KIIs): one each with the County Executive Committee representative or the county health director for medical services in each of the three counties where we will conduct our study, and one with the head of the division of NCDs at the MOH.

Methodology: Focus Group Discussions: Clinical staff will be recruited by identifying staff who care for patients with hypertension. Patients will be recruited from the health facilities participating in the study. We will work with the AMPATH leadership to identify local community members. FGD guides will be created specific to each target group, based on the COM-B constructs listed above (Table 1). Additionally, the FGDs of the clinical staff will assess organizational readiness for change (change efficacy, change commitment, and organizational context)<sup>134</sup> to implement a new multi-level strategy. Each guide will be pilot-tested on three individuals (male, female, and clinician) and revised accordingly. A trained moderator will lead each FGD and facilitate the discussion, <sup>135</sup> with an observer and a note-taker present. Each FGD will last approximately 60 to 90 minutes and will be audio-recorded. We will encourage interactions between and among group members <sup>136</sup> employing participatory techniques that elicit emotional elements and promote group interactions. <sup>137-139</sup> After each FGD, the facilitators will conduct a debriefing session to summarize findings, compare impressions, identify procedural problems, and develop plans for future FGDs

Key Informant Interviews (KIIs): The four key informants will be approached and recruited in collaboration with AMPATH CDM who have existing relationships with policymakers at both the national and county level. A trained research assistant will conduct each of the KIIs. Each KII will last approximately 30-45 minutes and will be audio-recorded. We will prepare and pilot-test an interview guide in a similar manner as above and revise it accordingly. In addition to asking about facilitators, barriers and contextual factors that may impact the strategy, the KIIs will also assess governmental readiness for change to implementing a new multi-level strategy. <sup>134</sup> For all qualitative sessions, a transport allowance and refreshments will be provided to participants.

Focus Group Discussions and Key Informant Interviews will be conducted in-person by the Principal Investigator (PI), Dr. Rajesh Vedanthan, or designated research team members, assisted by an interpreter. The study team will adhere to the COVID-19 regulations during the interviews including social distancing, wearing masks throughout the interviews, as well as sanitize and ensuring proper aeration. During the interview, the investigators will ask questions regarding incorporating health IT and peer delivery for improving medication adherence and control of blood pressure among hypertensive patients in PT4A participating communities.

Outcomes and Analysis: All FGDs and KII audio-recordings will be transcribed and translated into English by the research team, and all translated interviews will be double-checked for accuracy. We will perform content analysis of the transcripts and notes using NVIVO software. Specific quotations, group interactions, and observations will be assigned codes based on content. Two co-ls will code two transcripts independently, after which they will compare codes, arrive at consensus, and develop a coding list with definitions for the remaining transcripts. In order to assess inter-coder reliability, we will randomly select 10% of transcribed pages to be coded by two co-ls, and the Kappa-statistic will be calculated. Discrepancies will be adjudicated by a third qualitative research co-l. We will then search the remaining transcripts for the following deductive (a priori) codes: (a) perception of adherence to hypertension medication; (b) perception of HIT; (c) perceptions regarding the role of social support; (d) perception of peer delivery; and (e) factors that may impact the success of the PT4A strategy. Significant inductive

(emerging) codes will also be identified, assessing for differences by sex. Coded items will be grouped into a hierarchical, branching structure in which broad concepts are first identified. Then themes and interpretive ideas emerging from those constructs are labeled using constant comparison techniques, and subsequently synthesized using matrices structured by the main themes of the analysis. Had Findings from the FGDs and KIIs will inform the HCD strategy refinement (Sub-Aim 1.1).

<u>Limitations and Alternative Strategies</u>: We may have trouble recruiting for the FGDs. To mitigate this, we will adhere to the principles of community engagement as described above, and hold sensitization sessions among potential participants. Given our success recruiting for similar research recently, <sup>91,109</sup> we do not anticipate that this will be a significant issue. It is also possible to assess for these factors using a more quantitative approach. However, using the proposed type of qualitative methods, our team has successfully uncovered novel factors that have informed and impacted the implementation of previous strategies. <sup>91,143,144</sup> It is possible that we will identify factors that are not aligned with the planned components of the PT4A strategy; in this scenario, we will incorporate those factors into the human-centered design approach described in Aim 2.

# Aim 2: Use a human-centered design approach to refine and adapt the PT4A strategy (to be implemented following completion of Aim 1 activities)

We will pursue a participatory, iterative design process 122,123,145 and assemble a human centered design (HCD) team consisting of individuals representing stakeholder groups: research team, clinicians, pharmacists, peers, and patients with hypertension, informatics staff, and other providers involved in hypertension care. The design process will involve three phases: brainstorming, conceptualization, and creation. During <u>brainstorming</u>, the facilitator will review relevant information on adherence to hypertension medications, findings from Aim 1, and the PT4A prototype core principles and characteristics. In the <u>conceptualization</u> phase, the team will evaluate advantages and disadvantages of ideas resulting from brainstorming, and arrive at consensus regarding importance, feasibility, and congruence to the PT4A strategy goals, 146,147 in order to more concretely refine the strategy. In the <u>creation</u> phase, we will develop the refined PT4A strategy. Educational (for patients) and training (for peers) materials will be developed in English, Kiswahili, and other local languages as appropriate, using standard approaches to translation and back-translation.

Core components of the PT4A strategy will include a HIT component and a peer delivery component. Prototype characteristics of each are described as follows (Figure 3).

Health Information Technology: All of the HIT components will build upon, and be aligned with, the AMPATH Informatics infrastructure that has been established. We are working with leadership of the AMPATH Informatics program to ensure full alignment. Our PT4A intervention will augment AMRS to support peer-based delivery in four ways: 1) decision support and tailored adherence counselling: provide a patient-level and historical adherence summary that includes pill count, self-report, and clinical data synced with AMRS to generate tailored adherence counselling; 2) teleconsultation: facilitate teleconsultation via text or phone call between peers and clinicians; 3) tracking and accountability: provide timely prompts to peers when refills are near due, and capture participant signature to confirm receipt of medications to improve accountability; and 4) analytics:



patient-level medication use analytics to predict future stock requirements for pharmacy supply chain. The specific design and implementation of the above will be iteratively improved via the participatory design process, as described in Sub-Aim 1.1. Each peer will be equipped with a tablet loaded with the AMRS-POC software and specific encounter forms and other features associated with the HIT component of the PT4A intervention. A Programmer will be hired as part of the Research staff, in coordination with the AMPATH informatics Program and approval by the Moi Research and Sponsored Projects Office and they will provide

technical support and training for the peers.

Peer Delivery: This component will involve trained and paid peer-delivery agents who will cover a prescribed catchment area associated with each health facility in the intervention arm. Peers will play three roles: 1) Drug delivery: peers will deliver medication refills to the patient at a convenient location and time. Upon enrollment, clinical data from the AMRS, including the participant's current prescription and the next refill date, will be sent by AMRS to the pharmacy staff, in order for them to package the medication. Each patient's prescriptions will be individually packed in standard manufacturer-issued blister packs, which will be packaged in single-seal bags to prevent pilferage. A prompt will also be sent by AMRS to the peer, who will confirm with the patient delivery details (which drugs, quantity, location, date, and time for delivery). The peer will pick up the medication package from the pharmacy at the health facility and then deliver the medication to the patient, who will confirm receipt by digitally signing on the HIT tool. The peer will then request the next installment of medications from the pharmacy (via AMRS), accounting for any pills that the patient did not consume and are remaining in the blister pack. The peer will continue this cycle of medication delivery until the patient returns to the health facility for a follow-up clinic visit, when a new prescription will be issued by the clinician to the patient. The peer will then start a new prescription refill cycle for the patient. 2) Psychosocial support and adherence counseling: leveraging the peer-patient relationship, 148 and using the HIT-generated adherence data, the peer will provide adherence counseling and psychosocial support to patients at the time of medication delivery to address individual-level adherence barriers and any new issues that may have been discovered during Aim 1 activities. Peers will be trained in motivational interviewing, health coaching, and psychosocial support. 149 3) Enhance patient activation: peers will use health coaching strategies to address concerns regarding medications, hypertension and other NCDs, and relationship with clinicians, thereby enhancing patient activation. Training, mentorship, supervision and monitoring of clinicians and peers on clinical content will be performed by the clinician investigators on the study who are qualified to do so,

| complemented by the standard CDM training that is organized by Cians. Research assistant led training and supervision of peers will lated SOPs and other research content. | CDM leadership and clini-<br>l be limited to research re- |
|---|---|
| PT4A Protocol 1.4 23 <sup>rd</sup> November, 2022 | Page <b>17</b> of <b>86</b> |

### Sub Aim 2.1: Evaluate The Intervention For Acceptability And Appropriateness.

This will be implemented following completion of Aim 2 activities and analysis Sub Aim 2.2: Conduct A Pilot of the Intervention and Evaluate Feasibility.

We will also conduct a pilot of the strategy for up to 1-year and conduct further FGDs to evaluate feasibility. We will select three pilot health facilities, one from each county. We will hire one peer delivery agent per facility, train them in core roles and responsibilities, and equip them with

| Table 3: Accepta | Table 3: Acceptability, Appropriateness, and Feasibility of the PT4A Intervention |
|---|---|
| | Outcomes |
| Acceptability | Satisfaction with the proposed intervention design |
| /tooopiasiiity | Expressed interest or intention to participate |
| Appropriateness | Perceived relevance of intervention to address adherence |
| Appropriateriess | Perceived fit w ithin existing community and clinical infrastructure |
| Face ibility | Anticipated success of implementing intervention in this setting |
| Feasibility | Perceived ease of implementing the intervention |

tablets. Each peer will be stationed at a specific health facility and will be able to communicate directly with the clinicians, pharmacy staff, and patients. To maintain patient confidentiality, all research

staff and peers will receive study specific training on the need to at all times maintain participant confidentiality, in addition to receiving training in good clinical practice (GCP) and human subjects' protection (HSP) training. The HIT platform builds on the AMPATH OpenMRS system which encompasses patient data protection measures such as restricted access to authorized users only, which will further maintain patient confidentiality. We will recruit up to 100 patients from among these three facilities, targeting an equal number per county. In case there is a report of an adverse reaction to medications or new symptom by the participant to the peer during the pilot phase of the study, all peer navigators will be guided by a decision support system built into the HIT that will require the prompt notification of one of the two local pharmacist investigators in the study, as well as the patient's clinician. The peer will contact directly both the pharmacist investigator(s) and the appropriate clinician. Swift action will be taken based on the advisement of the clinician. Inclusion criteria will include age greater than 18 years, and currently enrolled in the AMPATH CDM program. Exclusion criteria will include acute illness requiring immediate medical attention, terminal illness, or inability to provide informed consent.

We will collect data through a survey on process and implementation measures such as completeness of the peer delivery, satisfaction of the patients, patient activation, and fidelity of delivery strategy. We will conduct FGDs with patients and clinicians then conduct KII (Key informant interviews) with the peer delivery agents, focusing on contextual issues impacting implementation, suggestions for modifications, and concepts of feasibility (Table 3). The target group size for the FGDs is 6-10 participants but If there are insufficient numbers, we will accommodate a smaller size. FGD transcripts, data management, and analysis will be performed as described above. We have used this approach previously with success. 80,91,112,150

We will evaluate the impact of the pilot on absolute mean change in SBP and medication adherence from baseline to up to 1 year. The primary adherence outcome is the pill count adherence ratio, 151 which is the proportion of prescribed doses taken over a 1-month time period, assessed at the end of the pilot. The primary implementation outcome is fidelity, measured as quantity and quality of intervention delivery as intended, 152 comprised of three components: confirmed medication delivery documented by patient e-signature, peer completion of the HIT form, and quality of data entry into the HIT form.

We will also create a retrospective comparator group of CDM patients, by querying AMRS, matched by sex, age, location and by initial blood pressure level. We will use their recorded blood pressure over time and compare the 3, month, 6 month and 1 year change in blood pressure to those of the patients receiving the PT4A intervention to evaluate the magnitude and variance of the intervention effects.

### Rigor and Reproducibility

In addition to the rigorous study design described above, as well as the <u>consideration of relevant biological variables including sex</u>, we will create a data archive that will contain raw study data (no personal identifiers). This will be available to other investigators upon formal request made to the AMPATH Research Manager, following the publication of the primary analyses of the project, and after the data have been appropriately checked, cleaned and de-identified. The archive will reside on a server for which appropriate firewalls and other forms of data protection will be installed for maximum security. Prospective users will complete an application for use of the data, which will include queries about the users' project hypotheses and proposed analyses. All NIH regulations and restrictions as well as HIPAA Security Rules regarding personal health information will be observed.

### Study Procedures, Materials, and Potential Risks

Aim 1: Qualitative data will not contain any patient identifiers. These data include transcripts of FGDs and KIIs, and observation notes. FGDs and KIIs will be digitally audio-recorded and uploaded with a coded identification number (no identifying names) as an audio file to an electronically secure database on a password-protected computer. These research data will be stored in a password-protected electronically secure database on a password-protected computer that will be known only to key research team members and the Study Coordinator. Once uploaded to the electronically secure database, the data will be deleted from the digital recording device. Any documents containing identifying information and consent documentation will be separated and added to the site's secure storage locker. Electronically captured data will transfer to the research database at the time of entry into the handheld device through a secure connection tunnel. All data on mobile devices will be encrypted and stored on the device's internal memory. All paper data collection forms will be reviewed by the Study Coordinator and Data Manager for completeness. Once validated, any sheets containing directly identifiable information and consent documentation will be separated and added to the site's secure storage locker. The remaining, de-identified pages will then be placed in a separate storage locker prior to data entry. Only key investigators and study personnel will have access to individually identifiable private information about human subjects. Transcription of the audio files will occur in Kenya. These transcripts will also be stored in an electronically secure database on a password-protected computer.

Aim 2, Sub-Aim 2.1 and Sub-Aim 2.2: All clinical patient-level data will be entered into the AM-PATH Medical Record System (AMRS) as per AMPATH's standard operating procedures. A separate, password-protected research database will retrieve data from AMRS via access that will be controlled through user authentication. All data collected on paper forms will be transferred to the password-protected REDCap research database hosted by Moi University, using double data entry. Electronically captured data will be collected using the REDCap Mobile App, which enables offline data collection, then transferred to the password-protected REDCap research database through a secure connection tunnel. All data on mobile devices will be encrypted and stored on the device's internal memory. All paper data collection forms will be reviewed by the Study Coordinator and Data Manager for completeness and the presence of prespecified "danger" values. Once validated, any sheets containing directly identifiable information and consent documentation will be separated and added to the site's secure storage locker. The remaining, de-identified pages will then be placed in a separate storage locker prior to data entry. Only key investigators and study personnel will have access to individually identifiable

private information about human subjects. Qualitative data will be collected and handled in the same manner as Aim 1 above.

All research activities will be performed by CITI-certified research staff members. All data will be stored on dedicated, password-protected computers. Any data stored on portable media will be PGP-encrypted, in order to ensure security of the data. Paper forms will be stored for the duration of the study, and for one year following in order to allow verification of any data as needed for reporting and publication purposes. The paper forms will then be shredded. The electronic data with a coded identification number only (and no identifying names) may be kept indefinitely, in a secure manner as described above. Many of the questions used in this study carry a minimal risk of harm. Some of the questions in the focus group discussions, and interviews may be personal and may be considered sensitive or embarrassing. However, the project personnel will take measures to ensure that each subject's confidential information is secure and cannot be linked back to one's identity by anyone not involved in the study. Furthermore, there could be personal psychological stress related to a newly diagnosed health condition.

### **Known Potential Benefits**

The benefits to the study participants are two-fold. First, the information and data collected in Aim 1 will impact the implementation of strategies which enhance the adherence to hypertension medications and we will be able to modify its implementation based on the results of the research. Thus, the results of the research have the potential to decrease the cardiovascular risk, morbidity and mortality associated with elevated blood pressure. In addition, the cluster randomized trial, multiple-criteria decision analysis, and spatial analysis results will reveal important information that will benefit the stakeholders and subjects involved in the research, as well as to other individuals not directly involved in the research. We feel strongly that the benefits of such knowledge and the potential impact on the implementation of AMPATH's chronic disease management program greatly outweigh the minimal risks of the research procedures as described in the Research Strategy.

The knowledge gained from this study will also yield a direct benefit to the communities residing in Bungoma, Trans Nzoia, and Uasin Gishu Counties due to the direct applicability of the results to program implementation. In addition, other clinical sites within the AMPATH network will also benefit from the results of this research. Finally, other resource-poor communities in low-, middle, and high-income countries may benefit from the results and insights generated from this project.

In sum, we believe that this project involves minimal to low risk to the research subjects. Research subjects themselves stand to benefit substantially from the research activities. In addition, the benefit of the information obtained and disseminated to the study population as well as the greater population of Kenya, and its use to design scalable medication adherence interventions for chronic disease management, far outweigh the risks associated with this study. The projects expected benefits far exceed the expected risks, and therefore has a very low risk-benefit ratio.

### ASSESSMENT OF POTENTIAL RISKS AND BENEFITS

# Adequacy of Protection Against Risks A. Informed Consent and Assent

The study team will consist of local personnel and individuals from western Kenya who are familiar with the region. With the support of AMPATH and community leadership, the key investigators and Study Coordinator from MTRH will approach the subjects involved in Aim 1 in-person. Written

consent will be obtained from each individual. Consent forms will standardize the description of the study and will be given to each subject. For Aim 1, activities requiring a consent form are the key informant interviews and focus group discussions. At the end of the subject's reading, the interpreter will ask the subject if s/he has any questions. Study candidates will be provided information in terms that they can fully understand, not exerting any overt or covert coercion. A consent document will be used that is written and explained in the language that the potential subject understands (Kiswahili or English). Extreme care will be taken to fully explain the benefits and risks of the research before consent is obtained. The consent forms will be written in lay terminology at approximately 6th grade level. For Aim 1, the study subjects will provide written informed consent prior to any focus group discussion or key informant interview.

For Aim 2, the clinician will invite AMPATH CDM Program patients with uncontrolled hypertension and who are eligible for the study from the health facility to enroll in the study on the day of their routine clinic visit. On that day, research team members will describe the research study and the study protocol, and ensure the patient meets eligibility criteria. For patients randomized to the PT4A intervention arm, participants of will be informed the Health Information Technology (HIT) functionality and the availability of peer delivery agents who can deliver the medications to them. As above, extreme care will be taken to fully explain the benefits and risks of the research study, before consent is obtained. Written informed consent will be obtained from all participants. For Aim 2, activities requiring a consent form are the human-centered design FGD and the human-centered design survey. For Aim 2.1, a consent form will be developed and implemented to obtain written informed consent to participate in the FGD. Finally, for Aim 2.2, consent forms will be developed and implemented to obtain written informed consent in the Aim 2.2 FGD and participation in the pilot study. The consent forms will be written in lay terminology at approximately 6th grade level. For FGDs, written informed consent will be obtained in the same manner as above.

Individuals will be free to refuse to participate in the study at any time during the period of the study. A refusal will not impact the health care available to the individual in any manner. Access to care will not be impacted in any manner by an individual's decision to opt out of this research project.

AMPATH's Chronic Disease Management program in western Kenya provides clinical care for diabetes and hypertension using a robust and evidence-based clinical protocol, and is available at the rural health facilities (all government of Kenya primary care facilities) in this region. This care program includes facility-based testing and counseling, referral to the nearest appropriate health facility, clinical care at the health facility, and follow-up as required. All of the nurses and clinical officers who staff the chronic disease management program at the health centers and rural dispensaries have been trained in hypertension management according to the AMPATH protocol. Both the management protocol and the chronic disease management trainings have been developed jointly with the Ministry of Health and the District Health Management Team (DHMT) (Government of Kenya). In addition to an initial training workshop, continuing medical education sessions are organized every quarter during which hypertension and other topics are covered. Refresher trainings are also planned on an annual basis in order to update and assess nurses' knowledge and practices regarding hypertension management. Finally, AMPATH has used novel and innovative smartphone technology to create a clinical decision support and record-keeping system for the clinicians at the health facilities, in order to ensure that the standard-of-care AMPATH hypertension management protocol is adhered to by the practitioners. All individuals with hypertension or suspected hypertension are provided care in these clinical settings. In addition to AMPATH CDM Program described above, clinical care is available at mission hospitals, private clinics, and referral hospitals, and every individual will be informed of his/her option to receive care at any of these health facilities. All individuals will be able to attend any of these health facilities for care, and this will not be impacted in any manner by an individual's decision to opt out of this research project. This will be made clear during the informed consent process.

### B. Protections Against Risk

The following principles and procedures for data collection will be followed at the research site in order to minimize risk and protect confidentiality:

- Data will be collected on coded forms, which do not include other personal identifiers.
- Only the tracking form will have the participant's name and identifiable information.
- Study records will be stored in locked cabinets in a locked room only accessible by key staff at MTRH in Eldoret, Kenya.
- Only the study personnel will have access to the data and the codes.
- All computerized information will be protected by access codes known only to key investigators and certain designated staff members.
- No data will be published with participant names.
- Data that are contained on a digital audio recording device will be PGP-encrypted and the only identifying information captured during the recording will be the recording of the participants' voices.

\_

- All staff members will be trained to keep participants' information confidential, and will be informed of the penalty for breach of confidentiality.
- Any data accessed by NYUGSoM study personnel will be viewed and stored only on MCIT-approved computers and software.

The consent form signed by the participant will provide written assurance that all individual data collected in the study will be kept confidential to the extent provided by the Privacy Act of 1974. AMPATH will provide file security so that confidential data are not released. Specifically, participants will be informed that: (1) the only people who will know that they are research participants are members of the research team and, if appropriate, their physicians or health care providers; (2) no individual identifying information about them will be disclosed to others, except if required by law; and (3) when the results of the study are published or discussed in

conferences, no information will be included that would reveal their identity. Any material that is digitally audio-recorded will be uploaded with a coded identification number (no identifying names) as an audio file to an electronically secure database. The only identifying information captured during the recording will be the recording of the participants' voices. These research data will be stored in an electronically secure database protected by password that will be known only to the Principal Investigator and the Study Coordinator. Once uploaded to the electronically secure database on a password-protected computer, the data will be deleted from the digital recording device to protect confidentiality and minimize the risk of breach of confidentiality. Transcription of the audio files will occur in Kenya by trained research team members who have undergone human subjects research training certification. Transcripts will not be shared with anyone outside of the study team.

All clinical patient-level data will be entered into the AMRS as per AMPATH's standard operating procedures. A separate, password-protected research database will retrieve data from AMRS via access that will be controlled through user authentication. All data collected on paper forms will be transferred to the research database using double data entry. Electronically captured data will transfer to the research database at the time of entry into the handheld device through a secure

connection tunnel. All data on mobile devices will be encrypted and stored on the device's internal memory.

All data management will be carried out by CITI-certified research staff members, and all data will be stored on dedicated, password-protected computers. Paper forms will be stored for the duration of the study, and for one year following in order to allow verification of any data as needed for reporting and publication purposes. The paper forms will then be shredded. The electronic data with a coded identification number only

(and no identifying names) may be kept indefinitely, in a secure manner as described above. Data containing residential locations/addresses (person-identifiers) are considered highly sensitive

To prevent inadvertent disclosures and ensure subject confidentiality, data entry and document storage for materials containing directly identifiable information (i.e., coversheets) will be handled by key investigators or the Study Coordinator. The Study Coordinator will be responsible for the secure handling and storage of survey documents for the duration of research activity at the study site. Once activities have been completed, coversheets will be collected and forwarded to the AMPATH research office, where they will be stored in a secure, locked cabinet within a secure, locked room. To minimize the number of people with access to the

coversheet data, all data entry will be conducted under the direct supervision of the Study Coordinator. Once identifiable data has been entered as described, paper-based documents will be returned to secure storage. Data collected in the study will be used for research purposes only. The results of this research project will be summarized for reports and may be summarized for presentation at meetings or in publications. No individual identities will be disclosed in any of these reports or presentations. Furthermore, No data will be reported on an individual basis; all findings will be presented in aggregate form.

We recognize that "macro-level" structural and environmental factors such as cost of medicines and poorly equipped health facilities may be more important than the peer delivery and HIT intervention. However, addressing these macro-level factors is integral to the AMPATH CDM Program's operations, which have already been universally applied to all of the rural health facilities throughout the research catchment area. For instance, AMPATH has established communitybased revolving fund pharmacies to ensure that there is adequate stock of the required medications in every rural health facility. The rural health facility committees described above are intimately involved with the establishment of these revolving fund pharmacies, in order to ensure community participation, ownership, and empowerment. The AMPATH pharmacy team has a pharmacy technician designated to supervise these revolving fund pharmacies and ensure accountability, proper storage and record-keeping. Likewise, the AMPATH CDM Program has equipped the rural health facilities with blood pressure machines, filing cabinets, desks, and other infrastructure to facilitate the clinical care program. In addition, the CDM program has consciously chosen to implement the clinical care program in the rural health facilities precisely because of proximity to the local communities, villages, and households. Moreover, as described above, AM-PATH has developed a training curriculum jointly with the MOH and the DHMT that addresses both the theoretical and practical aspects of diabetes and hypertension management. Combined with the clinical decision support, AMRS, mentorship, and supervision described above, AMPATH is implementing comprehensive strategies to optimize the human resources dedicated to hypertension management in this region. Finally, the AMPATH Safety Net Program is actively engaged in income-generating and financial security activities for the communities of western Kenya, in order to address the economic situation confronted by those populations. We feel that AMPATH's efforts to address these macro-level factors will both address human subjects concerns, as well as support the implementation of the intervention strategy described in the grant application.



# **MILESTONES** The milestones to be achieved for this portion of the project are listed in Table 4, along with details of each milestone's objectives, activity, target completion date, performance goal and metric, and anticipated challenges and mitigation strategies.

| | · | | | Complete = | | Dod: | | I |
|---|---|---|---|---|---|---|---|---|
| Aim | Milestone | Objective | Activity Develop study | Completion Date<br>(Month) | Performance Goal | Performance<br>Metric | Data Source | Anticipated Challenges and Potential Mitigation Challenge: Delays in coordinating SOPs across multiple |
| | | | protocols and<br>standard operating<br>procedures | M2 | 100% of SOPs<br>completed | # of SOPs started,<br>% finalized | Completed SOP document | regions <u>Mitigation:</u> Regular conference calls among investigators and research team members, clear and |
| | | 1. Develop<br>standard<br>operating<br>procedures and<br>study protocols | Develop data collection tools | M2 | 100% of data<br>collection tools<br>finalized by completion<br>date | # of data collection<br>tools initiated, %<br>successfully<br>completed | Data collection tools records | enforced deadlines. <u>Challenge</u> : Delays in creating uniform data collection tools across multiple regions <u>Mitigation</u> : Regular conference calls among investigators and research team members, rigorous pilot testing, consensus-building activities |
| Preparator | Preparatory Phase | | Receive IRB<br>approval | M2 | 100% protocol<br>approved by all parties<br>by completion date | % approval<br>received from<br>required parties | Finalized protocol<br>and supporting<br>documents | <u>Challenge</u> ; Delays in receiving approval for all updated study material<br><u>Mitigation</u> : team will work with the IRBs to streamline<br>approval process and will create a strategic plan to<br>ensure content quality and completeness |
| | | 2. Hire and train research team | Hire and training of staff | M3<br>(and ongoing as<br>new staff are hired) | 100% of staff hired<br>and trained by the<br>target completion date | # of new staff hired<br>and trained on<br>relevant study<br>methods | Sign-in sheets from trainings | <u>Challenge</u> : Unforeseen barriers related to HR hiring policies and procedures at Individual institutions Mitigation; Incorporate additional time for any additional unforeseen time barriers/institutions requirements that may delay onboarding and training of new staff, and adjust training schedule as necessary |
| | | | Obtain human<br>subjects training<br>certification | M3<br>(and ongoing as<br>new staff are hired) | 100% of staff have<br>completed human<br>subjects certification<br>by target completion<br>date | # staff that have<br>successfully<br>completed human<br>subjects training | Training record log<br>and documented<br>CITI certifications | <u>Challenge</u> : Human subjects research may take longer than anticipated.<br><u>Mitigation</u> : Research coordinator will create and review a training record log on a weekly basis of all research staff, and report to PI. |
| | | 1. Conduct | Develop and<br>conduct pre-tests of<br>qualitative interviews<br>and discussion<br>guides | M2 | 100% of all interview<br>and discussion guides<br>developed; & 100% of<br>all pre-tests conducted | # of interviews and discussion guides completed | Finalized interview<br>and discussion<br>guides | <u>Challenge</u> : Delays in creating uniform interview and discussion guides across multiple regions and countries <u>Mitigation</u> : Regular conference calls among investigators and research team members, rigorous pilot lesting, consensus-building activities |
| Aim 1 | | qualitative<br>interviews (Focus<br>Group<br>Discussions and<br>Key Informant<br>Interviews) | Conduct in-depth key<br>informant interviews<br>and FDG's | M5 | 100% of all interviews conducted | # of interviews conducted | Interviews | <u>Challenge:</u> All interviewees may not be available to be interviewed at scheduled times <u>Mitication:</u> Research coordinator and research assistants to schedule all participants with backup times scheduled as necessary |
| Identify micro- and<br>macro-level contextual<br>factors that might<br>influence the<br>implementation of the | Conduct a thorough<br>baseline contextual<br>assessment of<br>barriers and<br>facilitators for<br>implementing PT4A | | Transcribe and<br>translate interview<br>recordings | M5 | 100% of all interview<br>recordings transcribe<br>and translated | # of interviews<br>conducted,<br>translated, and<br>transcribed | Interview transcripts | <u>Challenges</u> ; Lengthy interview recordings; multiple<br>language translation required<br><u>Mitigation</u> . Allocate more time for transcription and<br>translation |
| PT4A strategy | implementing P14A | 2. Analyze | Create data analysis code book | M5 | 100% of code books<br>developed | # of code books<br>developed by<br>research team | Code books | Challenge: Difficulties in creating uniform coding scheme across multiple regions<br>Mitigation: Regular conference calls among qualitative investigators and analysts; Kappa statistic threshold |
| | | qualitative data | Code and analyze qualitative data | M6 | 100% of transcripts coded and analyzed | # transcripts coded<br>and analyzed | NVivo database | <u>Challenge</u> : Difficulties in harmonizing qualitative data<br>analysis across multiple regions<br>Mitigation: Documenting context-specific differences<br>that arise from the transcripts; ensure that qualitative<br>analytic learn consists of individuals representing all<br>regions and countries |
| | | 1. Human-<br>centered design<br>process | Conduct human-<br>centered design<br>process | M8 | 100% of<br>brainstorming,<br>conceptualization, and<br>creation of process<br>completed | # of HCD sessions completed | Sign-in sheets from sessions | Consumed: Uniously assembleing In-LD learn with addequate representation of all key stakeholders, and difficulty scheduling sufficient sessions based on stakeholder and project staff availability Mitcation; Incorporate additional time for any addition unforseesen time barriers/institutions requirements that may delay recruitment and implementations, and adjust schedule as necessary. |
| | Refine the peer<br>delivery and HIT<br>components | | Conduct FGDs with<br>patients, peers and<br>clinical staff | М9 | 100% of all interviews conducted | # of interviews conducted | Interviews | Challenge: All challenges from qualitative data collection from Alm 1 above will apply |
| Aim 2 Use a human-centered design approach to | | | Code and analyze qualitative data | M9 | 100% of transcripts coded and analyzed | # transcripts coded<br>and analyzed | NVivo database | Mitigation: All mitigation from qualitative data collection from Aim 1 above will apply, as appropriate |
| refine and adapt the<br>PT4A strategy | | | Pilot implementation | M11 | 100% of pilot activities implemented | # of patients who<br>were recruited and<br>received pilot<br>intervention | REDCap database | <u>Challences</u> : Unforeseen delays in county engagement; iower-than-anticipated enrollment <u>Mitication</u> : Community-based screening events, community entry, clinician engagement, approval from clinic and regional administrators |
| | | | Feasibility Testing | M12 | 100% of testing activities completed | # of FGDs<br>completed | Interviews | Challenge: All challenges from qualitative data collection from Aim 1 above will apply Mitigation: All mitigation from qualitative data collection from Aim 1 above will apply, as appropriate |
| | | | Analysis | M12 | 100% completion of<br>pilot data analysis | % of pilot data<br>analysis completed | Pilot data collected<br>on REDCap and<br>Nvivo | Challenge: Incomplete data from implementation phase<br>Mitigation: An algorithm that factors in missing data will<br>be developed prior to data collection |
| | Publications and abstracts related to the aims | Complete publications and abstracts related for Aims 1 and 2 | Prepare and submit<br>publications and<br>abstracts for peer<br>review to relevant<br>journals | M8, M12 | 100% of planned publications and abstracts submitted for review | # of abstracts and publications submitted | All data collected<br>and analyzed from<br>Aim 1&2 | Challence: delay in data collection and subsequent<br>analysis, thus preventing writing initiation and completion<br>Mitigation; incorporate additional time for completion of<br>writing of publications |
| | Research Products Subsequent R01 grant submission | | Rank potential study<br>regions according to<br>MCDA results and<br>other factors | M7 | 100% of study sites selected | # of clusters and<br>health facilities<br>selected | MCDA results; Aim<br>1 results | Challenges: All challenges from Aim 1 and Aim 2 Milestone activates below will apply; in addition, ranking might be subject to differential weighting. Milestone: All miligation strategies from Aim 1 and Aim Milestone: All miligation strategies from Aim 1 and Aim Zimilestone activities will apply; in addition, all investigators and relevant stakeholders if appropriate, will discuss and utilimately arrive at consensus for all study regions, study sites, and health facilities to be included in the subsequent RO1 |
| Research Products | | | Reach out to and<br>meet with key<br>stakeholders for<br>collaboration<br>(community<br>members, healthcare<br>workforce, and policy<br>makers) | M7 | 100% stakeholder<br>representation<br>reached from<br>community members<br>and leadership,<br>healthcare workforce,<br>and policy makers<br>across all enrollment<br>institutions | # of stakeholders<br>engaged at each<br>enrollment<br>institutions | Stakeholder<br>meetings and<br>signed letters of<br>engagement<br>agreements | <u>Challenge</u> : Difficulty of access due to the geographical location of facilities may be underestimated; stakeholders might be hesitant to collaborate Mittgatfor; A two-week buffer period will be provided for qualitative interviews with unforeseen access challenges |
| PT4A Pro | tocol 1.4 | subsequent R01 | Recruit and establish collaboration with baseline facilities | м <sup>7</sup><br>r, 2022 | 100% of facilities<br>recruited as baseline<br>study sites | # of facilities<br>recruited for<br>qualitative activities | Stakeholder<br>meetings and<br>signed letters of<br>engagement<br>agreement from<br>medical<br>superintendents | engage in community entry activities; attempt to align<br>project objectives with interests of all stakeholder parties. |
| | | 3. Submit R01 Grant<br>Application | Prepare and submit<br>R01 grant application | M7 | 100% of grant<br>submission activites<br>completed by<br>appropriate NIH<br>deadline | 1 R01 submitted grant | Analysis results from<br>Aim 1 and 2 as<br>available | Chollenge: delay in data collection and subsequent analysis, thus preventing possibility of completion of R01 application Mitigation: incorporate additional time for R01 grant application submission, based on NIH deadlines, if necessary |
| | | • | • | | | | • | * |

### **TABLE 4: PT4A MILESTONES1**

### Timeline

| | | | | | l | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | M1 | M2 | М3 | M4 | M5 | M6 | M7 | M8 | М9 | M10 | M11 | M12 |
| Preparatory Phase | | | | | | | | | | | | |
| Finalize protocol manuals | | | | | | | | | | | | |
| Finalize standard operating procedures | | | | | | | | | | | | |
| Develop data collection tools | | | | | | | | | | | | |
| IRB approval | | | | | | | | | | | | |
| Hire and train staff | | | | | | | | | | | | |
| Aim 1 | | | | | | | | | | | | |
| Focus Group Discussions | | | | | | | | | | | | |
| Key Informant Interviews | | | | | | | | | | | | |
| Analysis | | | | | | | | | | | | |
| Aim 2 | - | | | | | | | | | | | |
| Human-Centered Design Process | | | | | | | | | | | | |
| Sub-Aim 2.1 | | | | | | | | | | | | |
| Acceptability and Appropriateness Testing | | | | | | | | | | | | |
| Sub-Aim 2.2 | | | | | • | | | | | | | |
| Pilot Implementation | | | | | | | | | | | | |
| Feasibility Testing | | | | | | | | | | | | |
| Analysis | | | | | | | | | | | | |
| Research Products | | | | | | | | | | | | |
| Community dialogue and input | | * | * | * | | * | | * | | * | | * |
| International Advisory Committee Meetings | | | | х | | | | | | | | х |
| International Conferences | | | | | | | | § | | | | § |
| Publications | | | | | | | | ‡ | | | | ‡ |
| R01 Grant Application | | | | | | | Δ | | | | | |

### REFERENCES

- 1. GBD 2017: a fragile world. Lancet 2018;392:1683.
- 2. Global, regional, and national comparative risk assessment of 84 behavioural, environmental and occupational, and metabolic risks or clusters of risks for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet 2018;392:1923-94.
- 3. Forouzanfar MH, Liu P, Roth GA, et al. Global Burden of Hypertension and Systolic Blood Pressure of at Least 110 to 115 mm Hg, 1990-2015. JAMA: the journal of the American Medical Association 2017;317:165-82.
- 4. Huffman MD, Lloyd-Jones DM. Global burden of raised blood pressure: Coming into focus. JAMA: the journal of the American Medical Association 2017;317:142-3.
- 5. Chow CK, Teo KK, Rangarajan S, et al. Prevalence, awareness, treatment, and control of hypertension in rural and urban communities in high-, middle-, and low-income countries. JAMA 2013;310:959-68.
- 6. Irazola VE, Gutierrez L, Bloomfield G, et al. Hypertension Prevalence, Awareness, Treatment, and Control in Selected LMIC Communities: Results From the NHLBI/UHG Network of Centers of Excellence for Chronic Diseases. Global Heart 2016;11:47-59.
- 7. Mills KT, Bundy JD, Kelly TN, et al. Global Disparities of Hypertension Prevalence and Control: A Systematic Analysis of Population-Based Studies From 90 Countries. Circulation 2016;134:441-50.
- 8. Roth GA, Abate D, Abate KH, et al. Global, regional, and national age-sex-specific mortality for 282 causes of death in 195 countries and territories, 1980–2017: a systematic analysis for the Global Burden of Disease Study 2017. The Lancet 2018;392:1736-88.
- 9. Ettehad D, Emdin CA, Kiran A, et al. Blood pressure lowering for prevention of cardiovascular disease and death: a systematic review and meta-analysis. Lancet (London, England) 2016;387:957-67.
- 10. Thomopoulos C, Parati G, Zanchetti A. Effects of blood pressure lowering on outcome incidence in hypertension. 1. Overview, meta-analyses, and meta-regression analyses of randomized trials. Journal of hypertension 2014;32:2285-95.
- 11. Bundy JD, Li C, Stuchlik P, et al. Systolic Blood Pressure Reduction and Risk of Cardiovascular Disease and Mortality: A Systematic Review and Network Meta-analysis. JAMA Cardiol 2017;2:775-81.
- 12. Whelton PK. The elusiveness of population-wide high blood pressure control. Annual review of public health 2015;36:109-30.
- 13. Benjamin EJ, Blaha MJ, Chiuve SE, et al. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation 2017;135:e146-e603.
- 14. Stevens B, Verdian L, Pezzullo L, Tomlinson J, Zegenhagen S. The Economic Burden of Hypertension in Latin America. Value in Health 2016;19:A647-A8.
- 15. Wang G, Fang J, Ayala C. Hypertension-associated hospitalizations and costs in the United States, 1979-2006. Blood pressure 2014;23:126-33.
- 16. Gheorghe A, Griffiths U, Murphy A, Legido-Quigley H, Lamptey P, Perel P. The economic burden of cardiovascular disease and hypertension in low- and middle-income countries: a systematic review. BMC public health 2018;18:975.
- 17. Owolabi M, Olowoyo P, Miranda JJ, et al. Gaps in Hypertension Guidelines in Low- and Middle Income Versus High Income Countries: a Systematic Review. Hypertension (Dallas, Tex: 1979) 2016;68:1328-37.
- 18. De Geest S, Zullig LL, Dunbar-Jacob J, et al. ESPACOMP Medication Adherence Reporting Guideline (EMERGE). Annals of Internal Medicine 2018;169:30-5.

- 19. Perreault S, Dragomir A, White M, Lalonde L, Blais L, Bérard A. Better adherence to antihypertensive agents and risk reduction of chronic heart failure. Journal of internal medicine 2009;266:207-18.
- 20. Lowy A, Munk VC, Ong SH, et al. Effects on blood pressure and cardiovascular risk of variations in patients' adherence to prescribed antihypertensive drugs: role of duration of drug action. International journal of clinical practice 2011;65:41-53.
- 21. Du L, Cheng Z, Zhang Y, Li Y, Mei D. The impact of medication adherence on clinical outcomes of coronary artery disease: A meta-analysis. European journal of preventive cardiology 2017;24:962-70.
- 22. Simpson SH, Eurich DT, Majumdar SR, et al. A meta-analysis of the association between adherence to drug therapy and mortality. BMJ (Clinical research ed) 2006;333:15.
- 23. Kim S, Shin DW, Yun JM, et al. Medication Adherence and the Risk of Cardiovascular Mortality and Hospitalization Among Patients With Newly Prescribed Antihypertensive Medications. Hypertension 2016;67:506-12.
- 24. Chowdhury R, Khan H, Heydon E, et al. Adherence to cardiovascular therapy: a meta-analysis of prevalence and clinical consequences. European heart journal 2013;34:2940-8.
- 25. Roebuck MC, Liberman JN, Gemmill-Toyama M, Brennan TA. Medication adherence leads to lower health care use and costs despite increased drug spending. Health Affairs (Project Hope) 2011;30:91-9.
- 26. Peacock E, Krousel-Wood M. Adherence to Antihypertensive Therapy. The Medical clinics of North America 2017;101:229-45.
- 27. Vrijens B, Antoniou S, Burnier M, de la Sierra A, Volpe M. Current Situation of Medication Adherence in Hypertension. Front Pharmacol 2017;8.
- 28. De Geest S, Ruppar T, Berben L, Schönfeld S, Hill MN. Medication non-adherence as a critical factor in the management of presumed resistant hypertension: a narrative review. EuroIntervention 2014;9:1102-9.
- 29. Erdine S, Arslan E. Monitoring treatment adherence in hypertension. Curr Hypertens Rep 2013;15:269-72.
- 30. Kim S, Shin DW, Yun JM, et al. Medication Adherence and the Risk of Cardiovascular Mortality and Hospitalization Among Patients With Newly Prescribed Antihypertensive Medications. Hypertension (Dallas, Tex: 1979) 2016;67:506-12.
- 31. Whelton PK, Carey RM, Aronow WS, et al. 2017
- ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Journal of the American College of Cardiology 2018;71:e127-e248.
- 32. World Health O. WHO | ADHERENCE TO LONG-TERM THERAPIES: EVIDENCE FOR ACTION. WHO.
- 33. Abegaz TM, Shehab A, Gebreyohannes EA, Bhagavathula AS, Elnour AA. Nonadherence to antihypertensive drugs: A systematic review and meta-analysis. Medicine 2017;96:e5641.
- 34. Njuguna B, Vedanthan R. Find and Plug the Leak: Improving Adherence to Anti-Hypertensive Medicines: Editorial to: "Assessing Adherence to Antihypertensive Therapy in Primary Health Care in Namibia: Findings and Implications" by M.M. Nashilongo et al. Cardiovasc Drugs Ther 2017;31:485-7.
- 35. Tran DN, Njuguna B, Mercer T, et al. Ensuring Patient-Centered Access to Cardiovascular Disease Medicines in Low-Income and Middle-Income Countries Through Health-System Strengthening. Cardiology clinics 2017;35:125-34.
- 36. Burnier M, Egan BM. Adherence in Hypertension. Circulation research 2019;124:1124-40.

- 37. Macquart de Terline D, Kane A, Kramoh KE, et al. Factors associated with poor adherence to medication among hypertensive patients in twelve low and middle income Sub-Saharan countries. PLOS ONE 2019;14:e0219266.
- 38. Attaei MW, Khatib R, McKee M, et al. Availability and affordability of blood pressure-lowering medicines and the effect on blood pressure control in high-income, middle-income, and low-income countries: an analysis of the PURE study data. Lancet Public Health 2017;2:e411-e9.
- 39. Ambaw AD, Alemie GA, W/Yohannes SM, Mengesha ZB. Adherence to antihypertensive treatment and associated factors among patients on follow up at University of Gondar Hospital, Northwest Ethiopia. BMC public health 2012;12:282.
- 40. Khatib R, Schwalm J-D, Yusuf S, et al. Patient and Healthcare Provider Barriers to Hypertension Awareness, Treatment and Follow Up: A Systematic Review and Meta-Analysis of Qualitative and Quantitative Studies. PLoS One 2014;9.
- 41. Naanyu V, Vedanthan R, Kamano JH, et al. Barriers Influencing Linkage to Hypertension Care in Kenya: Qualitative Analysis from the LARK Hypertension Study. J Gen Intern Med 2016;31:304-14.
- 42. Rachlis B, Naanyu V, Wachira J, et al. Identifying common barriers and facilitators to linkage and retention in chronic disease care in western Kenya. BMC public health 2016;16:741.
- 43. Tamblyn R, Abrahamowicz M, Dauphinee D, et al. Influence of physicians' management and communication ability on patients' persistence with antihypertensive medication. Archives of internal medicine 2010;170:1064-72.
- 44. Schoenthaler A, Knafl GJ, Fiscella K, Ogedegbe G. Addressing the Social Needs of Hypertensive Patients: The Role of Patient-Provider Communication as a Predictor of Medication Adherence. Circulation Cardiovascular quality and outcomes 2017;10.
- 45. Schoenthaler A, Allegrante JP, Chaplin W, Ogedegbe G. The effect of patient-provider communication on medication adherence in hypertensive black patients: does race concordance matter? Ann Behav Med 2012;43:372-82.
- 46. Schoenthaler A, Montague E, Baier Manwell L, Brown R, Schwartz MD, Linzer M. Patient-physician racial/ethnic concordance and blood pressure control: the role of trust and medication adherence. Ethn Health 2014;19:565-78.
- 47. Berhe DF, Taxis K, Haaijer-Ruskamp FM, et al. Impact of adverse drug events and treatment satisfaction on patient adherence with antihypertensive medication a study in ambulatory patients. British journal of clinical pharmacology 2017;83:2107-17.
- 48. Lewis LM, Schoenthaler AM, Ogedegbe G. Patient factors, but not provider and health care system factors, predict medication adherence in hypertensive black men. J Clin Hypertens (Greenwich) 2012;14:250-5.
- 49. Fisher EB, Ballesteros J, Bhushan N, et al. Key Features Of Peer Support In Chronic Disease Prevention And Management. Health Affairs 2015;34:1523-30.
- 50. Enriquez M, Conn VS. Peers as Facilitators of Medication Adherence Interventions: A Review. J Prim Care Community Health 2016;7:44-55.
- 51. Haidari A, Moeini M, Khosravi A. The Impact of Peer Support Program on Adherence to the Treatment Regimen in Patients with Hypertension: A Randomized Clinical Trial Study. Iran J Nurs Midwifery Res 2017;22:427-30.
- 52. Nieuwlaat R, Wilczynski N, Navarro T, et al. Interventions for enhancing medication adherence. The Cochrane Database of Systematic Reviews 2014:CD000011.
- 53. Bosworth HB, Zullig LL, Mendys P, et al. Health Information Technology: Meaningful Use and Next Steps to Improving Electronic Facilitation of Medication Adherence. JMIR Med Inform 2016;4.

- 54. Dixon BE, Alzeer AH, Phillips EOK, Marrero DG. Integration of Provider, Pharmacy, and Patient-Reported Data to Improve Medication Adherence for Type 2 Diabetes: A Controlled Before-After Pilot Study. JMIR Med Inform 2016;4.
- 55. Dixon BE, Jabour AM, Phillips EOK, Marrero DG. An informatics approach to medication adherence assessment and improvement using clinical, billing, and patient-entered data. Journal of the American Medical Informatics Association: JAMIA 2014;21:517-21.
- 56. Bloomfield GS, Vedanthan R, Vasudevan L, Kithei A, Were M, Velazquez EJ. Mobile health for non-communicable diseases in Sub-Saharan Africa: a systematic review of the literature and strategic framework for research. Globalization and Health 2014;10:49.
- 57. Vedanthan R, Bernabe-Ortiz A, Herasme OI, et al. Innovative Approaches to Hypertension Control in Low- and Middle-Income Countries. Cardiology Clinics 2017;35:99-115.
- 58. World Health O. WHO | Impacts of e-health on the outcomes of care in low- and middle-income countries: where do we go from here? WHO.
- 59. Martin MY, Kim YI, Kratt P, et al. Medication adherence among rural, low-income hypertensive adults: a randomized trial of a multimedia community-based intervention. Am J Health Promot 2011;25:372-8.
- 60. Collaborators USBoD, Mokdad AH, Ballestros K, et al. The State of US Health, 1990-2016: Burden of Diseases, Injuries, and Risk Factors Among US States. JAMA: the journal of the American Medical Association 2018;319:1444-72.
- 61. Mainous AG, 3rd, King DE, Garr DR, Pearson WS. Race, rural residence, and control of diabetes and hypertension. Ann Fam Med 2004;2:563-8.
- 62. Kini V, Ho PM. Interventions to Improve Medication Adherence: A Review. JAMA: the journal of the American Medical Association 2018;320:2461-73.
- 63. Disease GBD, Injury I, Prevalence C. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet 2016;388:1545-602.
- 64. Zimmermann C, Swami N, Krzyzanowska M, et al. Perceptions of palliative care among patients with advanced cancer and their caregivers. CMAJ: Canadian Medical Association journal = journal de l'Association medicale canadienne 2016;188:E217-27.
- 65. Pino M, Parry R, Land V, Faull C, Feathers L, Seymour J. Engaging Terminally III Patients in End of Life Talk: How Experienced Palliative Medicine Doctors Navigate the Dilemma of Promoting Discussions about Dying. PLoS One 2016;11:e0156174.
- 66. Barasa FA, Vedanthan R, Pastakia SD, et al. Approaches to Sustainable Capacity Building for Cardiovascular Disease Care in Kenya. Cardiol Clin 2017;35:145-52.
- 67. Binanay CA, Akwanalo CO, Aruasa W, et al. Building Sustainable Capacity for Cardiovascular Care at a Public Hospital in Western Kenya. J Am Coll Cardiol 2015;66:2550-60.
- 68. Bloomfield GS, Xavier D, Belis D, et al. Training and Capacity Building in LMIC for Research in Heart and Lung Diseases: The NHLBI-UnitedHealth Global Health Centers of Excellence Program. Glob Heart 2016;11:17-25.
- 69. Truglio J, Graziano M, Vedanthan R, et al. Global health and primary care: increasing burden of chronic diseases and need for integrated training. Mt Sinai J Med 2012;79:464-74.
- 70. Miller ML, Karwa R, Schellhase EM, et al. Meeting the Needs of Underserved Patients in Western Kenya by Creating the Next Generation of Global Health Pharmacists. Am J Pharm Educ 2016;80:22.
- 71. Dodd R, Ramanathan S, Angell B, et al. Strengthening and measuring research impact in global health: lessons from applying the FAIT framework. Health Research Policy and Systems 2019;17:48.
- 72. Pastakia SD, Schellhase EM, Jakait B. Collaborative partnership for clinical pharmacy services in Kenya. American journal of health-system pharmacy: AJHP: official journal of the American Society of Health-System Pharmacists 2009;66:1386-90.

- 73. (Accessed July 3, 2019, at <a href="http://www.incap.int/ciipec/index.php/en/ciipecenglishv">http://www.incap.int/ciipec/index.php/en/ciipecenglishv</a>.)
- 74. Webster R, Parker G, Heritier S, et al. Strategic, Successful, and Sustained Synergy: The Global Alliance for Chronic Diseases Hypertension Program. Glob Heart 2019;14:391-4.
- 75. Yan LL, Vedanthan R, Mensah GA, et al. Developing the Core Pillars of Training Global Cardiovascular Health Researchers: Companionship, Light, and Fuel. Glob Heart 2019;14:387-9
- 76. Bazzano AN, Martin J, Hicks E, Faughnan M, Murphy L. Human-centred design in global health: A scoping review of applications and contexts. PLOS ONE 2017;12:e0186744.
  77. Ideo. Design Kit.
- 78. Vedanthan R, Kamano JH, Horowitz CR, et al. Nurse management of hypertension in rural western Kenya: implementation research to optimize delivery. Ann Glob Health 2014;80:5-12.
- 79. Vedanthan R, Kamano JH, Lee H, et al. Bridging Income Generation with Group Integrated Care for cardiovascular risk reduction: Rationale and design of the BIGPIC study. Am Heart J 2017;188:175-85.
- 80. Leung C, Naert M, Andama B, et al. A Human-Centered Design Approach to Develop a Microfinance and Group Medical Visit Model for Cardiovascular Risk Reduction in Western Kenya (BIGPIC Study) American Heart Association Annual Scientific Sessions; 2017 November; Anaheim, USA
- 81. Pillsbury MM, Mwangi E, Andesia J, et al. Human-centered design for global health implementation science: Lessons from the STRENGTHS study in western Kenya. Consortium of Universities for Global Health; 2020; Washington, DC.
- 82. Einterz RM, Kimaiyo S, Mengech HN, et al. Responding to the HIV pandemic: the power of an academic medical partnership. Acad Med 2007;82:812-8.
- 83. Mercer T, Gardner A, Andama B, et al. Leveraging the power of partnerships: spreading the vision for a population health care delivery model in western Kenya. Globalization and health 2018:14:44-.
- 84. Bloomfield GS, Kimaiyo S, Carter EJ, et al. Chronic noncommunicable cardiovascular and pulmonary disease in sub-Saharan Africa: an academic model for countering the epidemic. American heart journal 2011;161:842-7.
- 85. Vedanthan R, Kamano JH, Bloomfield GS, Manji I, Pastakia S, Kimaiyo SN. Engaging the Entire Care Cascade in Western Kenya: A Model to Achieve the Cardiovascular Disease Secondary Prevention Roadmap Goals. Glob Heart 2015;10:313-7.
- 86. Manji I, Manyara SM, Jakait B, et al. The Revolving Fund Pharmacy Model: backing up the Ministry of Health supply chain in western Kenya. International Journal of Pharmacy Practice 2016:24:358-66.
- 87. Pastakia S, Manji I, Mercer T. Noncommunicable Diseases And Essential Medicines. Health Affairs 2015;34:2003.
- 88. Tran DN, Manji I, Njuguna B, et al. Solving the problem of access to cardiovascular medicines: Revolving fund pharmacy models in rural western Kenya. BMJ Global Health 2020;In press.
- 89. Mamlin BW, Biondich PG, Wolfe BA, et al. Cooking Up An Open Source EMR For Developing Countries: OpenMRS A Recipe For Successful Collaboration. AMIA Annual Symposium Proceedings 2006;2006:529-33.
- 90. Pastakia SD, Karwa R, Kahn CB, Nyabundi JS. The evolution of diabetes care in the rural, resource-constrained setting of western Kenya. Ann Pharmacother 2011;45:721-6.
- 91. Naanyu V, Vedanthan R, Kamano JH, et al. Barriers Influencing Linkage to Hypertension Care in Kenya: Qualitative Analysis from the LARK Hypertension Study. Journal of general internal medicine 2016;31:304-14.

- 92. Lee DJ, Kamano JH, Tulienge D, et al. Estimating the Health Workforce Requirements for Hypertension Management in Rural Western Kenya. American Heart Association Annual Scientific Sessions. Orlando, USA2015.
- 93. Rachlis B, Karwa R, Chema C, et al. Targeted Spontaneous Reporting: Assessing Opportunities to Conduct Routine Pharmacovigilance for Antiretroviral Treatment on an International Scale. Drug safety 2016;39:959-76.
- 94. Karwa R, Maina M, Mercer T, et al. Leveraging peer-based support to facilitate HIV care in Kenya. PLoS Med 2017;14:e1002355.
- 95. Inui TS, Sidle JE, Nyandiko WM, et al. 'Triangulating' AMPATH: demonstration of a multiperspective strategic programme evaluation method. SAHARA J 2009;6:105-14.
- 96. Park PH, Wambui CK, Atieno S, et al. Improving Diabetes Management and Cardiovascular Risk Factors Through Peer-Led Self-management Support Groups in Western Kenya. Diabetes care 2015;38:e110-1.
- 97. Pastakia SD, Karwa R, Kahn CB, Nyabundi JS. The evolution of diabetes care in the rural, resource-constrained setting of western Kenya. The Annals of pharmacotherapy 2011;45:721-6.
- 98. Rajput ZA, Mbugua S, Amadi D, et al. Evaluation of an Android-based mHealth system for population surveillance in developing countries. J Am Med Inform Assoc 2012;19:655-9.
- 99. Vedanthan R, Blank E, Tuikong N, et al. Usability and feasibility of a tablet-based Decision-Support and Integrated Record-keeping (DESIRE) tool in the nurse management of hypertension in rural western Kenya. Int J Med Inform 2015;84:207-19.
- 100. Were MC, Kamano JH, Vedanthan R. Leveraging Digital Health for Global Chronic Diseases. Glob Heart 2016;11:459-62.
- 101.Engelgau MM, Sampson UK, Rabadan-Diehl C, et al. Tackling NCD in LMIC: Achievements and Lessons Learned From the NHLBI-UnitedHealth Global Health Centers of Excellence Program. Glob Heart 2016;11:5-15.
- 102. Siika AM, Rotich JK, Simiyu CJ, et al. An electronic medical record system for ambulatory care of HIV-infected patients in Kenya. Int J Med Inform 2005;74:345-55.
- 103. Tierney WM, Achieng M, Baker E, et al. Experience implementing electronic health records in three East African countries. Studies in health technology and informatics 2010;160:371-5.
- 104.Pastakia SD, Ali SM, Kamano JH, et al. Screening for diabetes and hypertension in a rural low income setting in western Kenya utilizing home-based and community-based strategies. Globalization and health 2013;9:21.
- 105. Pastakia SD, Manyara SM, Vedanthan R, et al. Impact of Bridging Income Generation with Group Integrated Care (BIGPIC) on Hypertension and Diabetes in Rural Western Kenya. Journal of general internal medicine 2017;32:540-8.
- 106.Peiris D, Thompson SR, Beratarrechea A, et al. Behaviour change strategies for reducing blood pressure-related disease burden: findings from a global implementation research programme. Implementation science: IS 2015;10:158.
- 107. Vedanthan R, Kamano JH, Horowitz CR, et al. Nurse management of hypertension in rural western Kenya: implementation research to optimize delivery. Annals of global health 2014;80:5-12.
- 108. Vedanthan R, Kamano JH, Naanyu V, et al. Optimizing linkage and retention to hypertension care in rural Kenya (LARK hypertension study): study protocol for a randomized controlled trial. Trials 2014;15:143.
- 109. Vedanthan R, Tuikong N, Kofler C, et al. Barriers and Facilitators to Nurse Management of Hypertension: A Qualitative Analysis from Western Kenya. Ethn Dis 2016;26:315-22.
- 110. Schwalm JD, McKee M, Huffman MD, Yusuf S. Resource Effective Strategies to Prevent and Treat Cardiovascular Disease. Circulation 2016;133:742-55.

- 111.Embleton L, Wachira J, Kamanda A, Naanyu V, Ayuku D, Braitstein P. Eating sweets without the wrapper: perceptions of HIV and sexually transmitted infections among street youth in western Kenya. Culture, health & sexuality 2016;18:337-48.
- 112. Embleton L, Ott MA, Wachira J, et al. Adapting ethical guidelines for adolescent health research to street-connected children and youth in low- and middle-income countries: a case study from western Kenya. BMC medical ethics 2015;16:89.
- 113. Wachira J, Kamanda A, Embleton L, et al. Initiation to street life: a qualitative examination of the physical, social, and psychological practices in becoming an accepted member of the street youth community in Western Kenya. BMC public health 2015;15:569.
- 114. Wachira J, Kamanda A, Embleton L, Naanyu V, Ayuku D, Braitstein P. 'Pregnancy Has Its Advantages': The Voices of Street Connected Children and Youth in Eldoret, Kenya. PLoS One 2016;11:e0150814.
- 115.Embleton L, Wachira J, Kamanda A, et al. "Once you join the streets you will have to do it": sexual practices of street children and youth in Uasin Gishu County, Kenya. Reproductive health 2015;12:106.
- 116. Naanyu V, Sidle JE, Frankel RM, Ayuku D, Nyandiko WM, Inui TS. Rooting inquiry in tradition: the health baraza as a tool for social research in Kenya. Qual Health Res 2011;21:14-26.
- 117. Naanyu V, Asirwa CF, Wachira J, et al. Lay perceptions of breast cancer in Western Kenya. World journal of clinical oncology 2015;6:147-55.
- 118. Naanyu V, Baliddawa J, Peca E, Karfakis J, Nyagoha N, Koech B. An examination of postpartum family planning in western Kenya: "I want to use contraception but I have not been told how to do so". African journal of reproductive health 2013;17:44-53.
- 119.Leatherman S, Metcalfe M, Geissler K, Dunford C. Integrating microfinance and health strategies: examining the evidence to inform policy and practice. Health policy and planning 2012;27:85-101.
- 120.Kamanda A, Embleton L, Ayuku D, et al. Harnessing the power of the grassroots to conduct public health research in sub-Saharan Africa: a case study from western Kenya in the adaptation of community-based participatory research (CBPR) approaches. BMC public health 2013;13:91.
- 121. Vreeman R, Kamaara E, Kamanda A, et al. A qualitative study using traditional community assemblies to investigate community perspectives on informed consent and research participation in western Kenya. BMC medical ethics 2012;13:23.
- 122.Amin R, St Pierre M, Ahmed A, Haq R. Integration of an Essential Services Package (ESP) in child and reproductive health and family planning with a micro-credit program for poor women: experience from a pilot project in rural Bangladesh. World Development 2001;29:1611-21.
- 123. Pronyk PM, Hargreaves JR, Kim JC, et al. Effect of a structural intervention for the prevention of intimate-partner violence and HIV in rural South Africa: a cluster randomised trial. Lancet 2006;368:1973-83.
- 124. Porter CM. Revisiting Precede—Proceed: A leading model for ecological and ethical health promotion. Health Education Journal 2016;75:753-64.
- 125. Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Medical care 2012;50:217-26.
- 126.Mercer T, Njuguna B, Bloomfield GS, et al. Strengthening Referral Networks for Management of Hypertension Across the Health System (STRENGTHS) in western Kenya: a study protocol of a cluster randomized trial. 5th Global Symposium on Health Systems Research. Liverpool, UK2018.

- 127. Paradis G, O'Loughlin J, Elliott M, et al. Coeur en sante St-Henri--a heart health promotion programme in a low income, low education neighbourhood in Montreal, Canada: theoretical model and early field experience. Journal of epidemiology and community health 1995;49:503-12.
- 128. Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci 2011;6:42.
- 129. Jackson C, Eliasson L, Barber N, Weinman J. Applying COM-B to medication adherence: a suggested framework for research and interventions. The European Health Psychologist 2014;16.
- 130.McEvoy CT, Moore SE, Appleton KM, et al. Development of a peer support intervention to encourage dietary behaviour change towards a Mediterranean diet in adults at high cardiovascular risk. BMC public health 2018;18:1194.
- 131.Phillips R, Copeland L, Grant A, et al. Development of a novel motivational interviewing (MI) informed peer-support intervention to support mothers to breastfeed for longer. BMC Pregnancy Childbirth 2018;18:90.
- 132. Crayton E, Wright AJ, Ashworth M. Improving medication adherence in stroke survivors: the intervention development process. BMC health services research 2018;18:772.
- 133. Aseyo RE, Mumma J, Scott K, et al. Realities and experiences of community health volunteers as agents for behaviour change: evidence from an informal urban settlement in Kisumu, Kenya. Hum Resour Health 2018;16:53.
- 134. Weiner BJ. A theory of organizational readiness for change. Implement Sci 2009;4:67.
- 135.Fedder DO, Chang RJ, Curry S, Nichols G. The effectiveness of a community health worker outreach program on healthcare utilization of west Baltimore City Medicaid patients with diabetes, with or without hypertension. Ethn Dis 2003;13:22-7.
- 136.Hill MN, Bone LR, Hilton SC, Roary MC, Kelen GD, Levine DM. A clinical trial to improve high blood pressure care in young urban black men: recruitment, follow-up, and outcomes. Am J Hypertens 1999;12:548-54.
- 137. Parsell G, Gibbs T, Bligh J. Three visual techniques to enhance interprofessional learning. Postgrad Med J 1998;74:387-90.
- 138. Parsell G, Spalding R, Bligh J. Shared goals, shared learning: evaluation of a multiprofessional course for undergraduate students. Med Educ 1998;32:304-11.
- 139. Stuttaford M, Bryanston C, Hundt GL, Connor M, Thorogood M, Tollman S. Use of applied theatre in health research dissemination and data validation: a pilot study from South Africa. Health (London, England: 1997) 2006;10:31-45.
- 140.Dodd R, Munck L. Dying for change: poor people's experience of health and ill-health: World Health Organization and World Bank; 2002.
- 141. Hsieh H-F, Shannon SE. Three Approaches to Qualitative Content Analysis. Qualitative Health Research 2005;15:1277-88.
- 142. Vaismoradi M, Jones J, Turunen H, Snelgrove S. Theme development in qualitative content analysis and thematic analysis. Journal of Nursing Education and Practice 2016;6:100-10.
- 143.Rusk A, Goodman C, Naanyu V, Koech B, Obala A, O'Meara WP. Expanding Access to Malaria Diagnosis through Retail Shops in Western Kenya: What Do Shop Workers Think? Malaria research and treatment 2013;2013:398143.
- 144. Douglas A, Rotich J, Kiptoo P, et al. Development and Validation of a Behavioral Assessment for Optimizing Linkage to Hypertension Care in Kenya: The LARK Study. American Public Health Association Annual Meeting. Chicago, USA. 2014.
- 145.Kim J, Ferrari G, Abramsky T, et al. Assessing the incremental effects of combining economic and health interventions: the IMAGE study in South Africa. Bulletin of the World Health Organization 2009;87:824-32.
- 146. Chen EK, Reid MC, Parker SJ, Pillemer K. Tailoring evidence-based interventions for new populations: a method for program adaptation through community engagement. Evaluation & the health professions 2013;36:73-92.
- 147. Weiner BJ, Lewis CC, Stanick C, et al. Psychometric assessment of three newly developed implementation outcome measures. Implementation Science 2017;12:108.
- 148. Funnell MM. Peer-based behavioural strategies to improve chronic disease self-management and clinical outcomes: evidence, logistics, evaluation considerations and needs for future research. Family Practice 2010;27:i17-22.
- 149. Ogedegbe G, Chaplin W, Schoenthaler A, et al. A practice-based trial of motivational interviewing and adherence in hypertensive African Americans. Am J Hypertens 2008;21:1137-43.
- 150. Sanders D, Haines A. Implementation research is needed to achieve international health goals. PLoS Med 2006;3:e186.

# APPENDIX A. PT4A AIM 2 STUDY PROTOCOL

<u>Project Title</u>: Human Centered Implementation Research for refining and adapting the Peers and Technology for Adherence, Access, Accountability and Analytics (PT4A) Strategy.

Abstract: Medication adherence is a much needed avenue of recourse in order to reduce cardiovascular disease (CVD) and death resulting from complications of high BP<sup>1-4</sup>. To address these hurdles, we hypothesize that the PT4A strategy, which has a component of peer delivery of medication and Health Information Technology, can be an effective implementation strategy to positively influence several micro- and macro-level factors leading to improved adherence to hypertension medications. In this study we will use the human centered design (HCD) approach to refine this proposed strategy. HCD is increasingly applied to implementation research, and it has successfully been used in previous studies<sup>7-8</sup>. This process starts with the people you are designing for and ends with new solutions that are tailor-made to suit their needs. It builds upon participatory action research, and our protocol includes: patients who are hypertensive, clinical teams providing care to the patients, and community members, who will provide insights on HTN management in a community setting. Initial stages usually revolve around immersion, observing, and contextual framing in which innovators immerse themselves with the problem and community. Subsequent stages may then focus on community brainstorming, modeling and prototyping, and implementation in community spaces. <sup>9</sup> The PT4A Strategy will undergo the following human-centered design processes: the Inspiration phase, Ideation phase, and Implementation phase. An HCD team consisting of individuals representing stakeholder groups: research team, clinicians, pharmacists, peers, patients with hypertension, informatics staff, and other providers involved in hypertension care will go through a participatory and iterative process to help in refining this implementation strategy.

In the Inspiration phase we will learn directly from the people we are designing for. In this case using qualitative research methods as described in Aim 1, we will conduct a thorough baseline contextual assessment of barriers and facilitators for implementing PT4A, and will gain a deeper understanding of the patients, community, and healthcare workers needs and opportunities for solutions. The interview questions employed participatory techniques that elicited emotional elements and promoted group interactions. <sup>10-12</sup>. The information that will form the guiding themes that will inform the PT4A strategy refinement include: (a) perception of adherence to hypertension medication, (b) perception of HIT, (c) perceptions regarding the role of social support, (d) perception of peer delivery, and (e) factors that may impact the success of the PT4A strategy.

We will explore insights into tangible ideas, divergence and convergence coming closer to the solution that can work best. It is the expectation that team members can have varying ideas when giving solutions but through the process we are able to get a solution that can work and is acceptable with many.

In the Ideation phase we will make sense of the information learned, identify opportunities for design, and prototype possible solutions. During this phase we will look at the actionable items around the core structure of using a peer to deliver medication and the use of the mobile device as a health information support tool.

In the Implementation phase we will bring the solution to life, and eventually, to implementation in the real world. Once the refined PT4A strategy model is developed, we will conduct o assess acceptability and appropriateness. Participants will be recruited through convenience sampling and will provide written informed consent. The initial prototype diagrams will convey key

PT4A Protocol 1.4 23<sup>rd</sup> November, 2022

features of the strategy to the participants and depicted use from the patient, clinician, and peer delivery agent perspectives.

#### **PARTICIPANTS**

A team consisting of individuals representing stakeholder groups (in total number 20): research team, clinicians, pharmacists, peers, patients with hypertension, informatics staff, and other providers involved in hypertension care will make up the design team. They will be recruited from across the three counties participating in the study. Participants will be reimbursed for their time, transportation and will be served a snack during design team meetings.

#### **METHODOLOGY:**

The design team (DT) will meet for a total of 6 meetings over the course of the process, in order to develop and iteratively adapt the integrated door to door peer delivery of medication and Health Information Technology (HIT) intervention.

**Preliminary Activities:** Baseline information will directly inform our design process. Data collected using qualitative methods that consist of key informant interviews and focus group discussions on the Micro and Macro level contextual factors (individual, family, clinician, health system) that might influence the implementation of the PT4A strategy will be presented before commencing our HCD design process; information on this process can be found in the parent study protocol.

**Baseline Technology:** All of the HIT components will build upon, and be aligned with, the AM-PATH Informatics infrastructure that has been established.

Our PT4A intervention will augment AMRS to support peer-based intervention in four ways:

- 1) <u>Decision support and tailored adherence counseling:</u> provide a patient-level and historical adherence summary that includes pill count, self-report, and clinical data synced with AMRS to generate tailored adherence counseling;
- 2) <u>Teleconsultation</u>: facilitate teleconsultation via text or phone call between the patients and clinicians, by the help of the peer.
- 3) <u>Tracking and accountability</u>: provide timely prompts to peers when refills are near due, and capture participant signature to confirm receipt of medications to improve accountability.
- 4) A<u>nalytics</u>: patient-level medication use analytics to predict future stock requirements for pharmacy supply chain. The specific design and implementation of the above will be iteratively improved via the participatory design process.

<u>Design Process Goals:</u> The Design Team will be asked to identify and prototype potential solutions to issues raised in the baseline needs and contextual assessment, in addition to the following 4 core elements of the integrated HIT, the door-to-door medication delivery, and peer support intervention:

#### **Design Team Meeting #1: Inspiration**

#### Session A:

- DT members will introduce themselves and review expectations for the design process, including the scope of work for the design team and the expected process to be followed during the design team, including the role of the research team in co-design and approval of the final intervention.
- PT4A research team members will introduce human-centered design methods through a presentation

PT4A Protocol 1.4 23<sup>rd</sup> November, 2022

• DT members will share their personal experiences with patient medication adherence challenges and support.

### Session B:

- PT4A research team will introduce findings from Aim 1 activities; the design team will
  compile salient and interesting insights from the following findings: (a) perception of adherence to hypertension medication; (b) perception of HIT; (c) perceptions regarding the
  role of social support; (d) perception of peer delivery; and (e) factors that may impact the
  success of the PT4A strategy and create post-it notes
- Notes will be posted on the walls and arranged into clusters based on topics and patterns, forming central themes

## **Expected outcomes:**

- Introduction and group logistics
- Understanding of the HCD process and definition of roles
- Creation of themes that we lead to development of insight statements.
- Start the synthesis process of ideation

# **Design Team Meeting #2: Brainstorming**

#### Session A:

- DT members will engage in icebreaker activities & review previous meeting discussions.
- PT4A STUDY research team will identify themes based on summary statements from DT Meeting #1
- DT will break into small groups and create "How might we..." questions to address summary statements (i.e. "How might peers best deliver the medication?")
- DT will select up to 5 HMW (How Might We) questions and post them on the wall

#### Session B:

- DT will break into small groups and brainstorm solutions to each problem in 15-minute rotations (i.e. "the peers delivering medication and offering psychosocial support")
- PT4A team will introduce baseline core functions for the peers as follows and address HWM around the following issues to be addressed.
  - 1) Drug delivery: peers will deliver medication refills to the patient at a convenient location and time.
  - 2) Confirmation of the medicine delivery with the patient delivery details (which drugs, quantity, location, date, and time for delivery).
  - 3) Psychosocial support and adherence counseling: leveraging the peer-patient relationship and using the HIT-generated adherence data, the peer will provide adherence counseling and psychosocial support to patients at the time of medication delivery to

address individual-level adherence barriers and any new issues that may have been discovered during Aim 1 activities.

Beyond the above, the DT may deliberate on additional functions for the peers, or introduce subfunctions within the above

# **Expected outcomes:**

Creation of insight statements that will lead to how might we questions

# **Design Team Meeting #3: Conceptualization**

#### Session A:

- DT members will engage in icebreaker activities & review previous meeting discussions.
- DT will discuss how might we question and propose each solution, evaluate advantages/disadvantages, and group similar ideas together
- DT will discuss the positive and negative effects of the proposed solutions.
- DT will vote to select up to 3 solution ideas for each HMW (How Might We) question
- DT will break into small groups and storyboard stakeholders' experience with this intervention using wall notes

#### Session B:

- DT will discuss each storyboard as a large group and select 1-2 solutions for each HMW question that will be prototyped during acceptability testing. If not already discussed, DT will address background logistics that underlie this integrated peer support intervention, including:
  - The peer role
    - How peers are recruited (Age, Gender, Education level)
    - Peer-patient relationship (Interpersonal skills)
    - The frequency of contact between the peer and the patients
    - The mechanism of contact with patients (SMS, phone, etc.)
    - The process of delivery of medication refills to the patient at a convenient location and time.
    - Confirmation of the medication delivery

## **Expected outcomes:**

Discuss the strongest solutions proposed

#### Design Team Meeting #4: Creation

#### Session A:

- DT members will engage in icebreaker activities & review previous meeting discussions
- DT members will discuss the solutions in detail and come up with models as to where we
  will refine the proposed intervention
- The research team will integrate selected solutions into a first-draft intervention model PT4A Protocol 1.4 23<sup>rd</sup> November, 2022

#### Session B:

- The draft interventional model will be presented and members will be asked to provide for any additional input they may have.
- DT will present intervention model to the study investigators, AMPATH Informatics team, and other key stakeholders
- Investigators will be invited to provide input and discuss intervention features with the DT

## **Expected outcomes:**

- Present final intervention model
- Finish creation of training materials

Throughout the process, the research team will develop training materials for providers and peers, data collection and encounter forms, and the questionnaires to be used during acceptability testing, PT4A research team members will maintain frequent and ongoing communication with the DT throughout the process. The PT4A research team and Informatics team will be responsible for ensuring that the DT proposes solutions that are compatible with existing technologic capabilities and feasible within the health system.

## **Outcomes and Analysis**

Throughout the DT meetings, a designated scribe will take detailed notes, photographs, and audio records to capture the design process and how each idea was developed. This data will be used as descriptive indicators of our design process and group participation. The DT will submit a first-draft model of the intervention to the investigators, the research team, and AMPATH Informatics team. This model will include the basic features of the intervention, detailed descriptions of the different roles involved, and a description of the patient, peer delivery agent and provider experience in a variety of scenarios. The research team and Informatics team will be responsible for creating the prototype of this model for acceptability testing.

#### Subaim 2.1: Evaluate the intervention for acceptability and appropriateness

After the PT4A model prototype is created we will evaluate how applicable and workable the core components of PT4A will be more so in terms of cost, complexity, usability, and value.

Participants (targeted number of 39 in total will be enrolled), this will include representatives of the end users of our product, which includes: hypertension patients (5 per site), clinicians (5 per site), pharmacy (1 per site) and peers (6 in total). Participants will be recruited through convenience sampling within the 3 counties where we will conduct the study. Participants will be reimbursed for time and travel through PT4A funds during those sessions.

#### Methods:

Participants will be recruited through convenience sampling and will provide written informed consent. We will conduct surveys in three counties with a similar distribution of participants to gauge PT4A Protocol 1.4 23<sup>rd</sup> November, 2022

perspectives from various stakeholders in the model; this will include patients, peers, and clinical staff. Initial prototype diagrams will be shared with the group and presented from the perspective of each type of stakeholder to fully inform them of their role within the model. A structured questionnaire will be used to elicit constructive feedback from the group.

## **Outcomes and Analysis:**

Statistical Analysis will include descriptive statistics of outcomes of interest including:

1) Satisfaction with the proposed intervention design, 2) perceived appropriateness, 3) fit within existing community and clinical infrastructures, 4) perceived positive or negative effects, 5) expressed interest or intention to participate, 6) perceived relevance to address adherence to medication, 7) barriers to implementation within existing community and clinical infrastructure, 8) ease of implementing this intervention. At the conclusion of this analysis, the design team will meet to review these outcomes and refine the intervention model as necessary to enhance acceptability.

## <u>Design Team Meeting #5: Iteration 1</u>

#### Session A:

- DT members will engage in icebreaker activities and review the last meeting discussions
- The PT4A research team will present and discuss findings from acceptability and appropriateness testing
- DT will group issues raised from the interview surveys into themes and propose intervention updates

### Session B:

- DT will create an updated intervention model and submit this to the study investigators, research team, and Informatics team
- DT will be divided into two groups and participate in FGDs to evaluate their experience during the HCD process

#### Subaim 2.2: Conduct a pilot of the intervention and evaluate feasibility

#### Participants:

Three health facilities will participate in the pilot (one from each county involved in the study). One peer delivery agent will be hired per facility and will be in close contact with clinicians, pharmacy staff, and patients at each health facility. The study will include all who are involved in the care for these patients and we target to enroll a total of up to 100 patients in this phase. Ten patients per facility.

#### Inclusion criteria

- Greater than 18 years of age.
- Currently enrolled in an AMPATH CDM Program

## Exclusion criteria

- Acute illness requiring immediate medical attention
- Terminal illness
- Inability to provide informed consent

#### Methods:

PT4A Protocol 1.4 23<sup>rd</sup> November, 2022

The pilot study will be conducted over a 3-month period. Peers will be paid through the PT4A funds. After recruitment and hiring, they will be on-boarded through a week-long training that will cover: i) basic training on hypertension care, ii) use of the PT4A HIT tool to ensure proper documentation of medication pick-up, medication delivery, and peer-patient encounter documentation; iii) providing psychosocial support for hypertensive patients aimed at supporting medication adherence and promoting patient activation. Peers will use the AMRS system (peers will have access to a tablet with access to the HIT/AMRS system, and technological support will be provided by research and the Ampath informatics team) to request a prescription for a patient in the provider catchment. The AMRS system will send the prescription from the healthcare provider to the pharmacy that covers that network. The pharmacy will prepare individually sealed blister bags in individual single seal bags to lower pilferage. Once packaging is complete, the AMRS system will send a message to the peer with the name, date/time of delivery, location, type of drug, and quantity to ensure the right medication is picked up at the right time. The peer will pick up the prescription and then deliver the medication to the patient, confirming receipt by getting a signature from the patient on the HIT tool. The peer will then request the next installment of medications through the AMRS system, taking into account any pills not consumed (remaining in the blister pack). This cycle will repeat until the patient has to see the clinician again, where the clinician will provide a new prescription. During these deliveries, peers will leverage adherence data to support patients and address any barriers to medication adherence. The overall goal of this psychosocial support will be increasing patient activation.

### Outcomes and Analysis:

We will collect data on implementation such as completeness of the peer delivery, satisfaction of the patients, patient activation, and fidelity of delivery strategy. Patient satisfaction will be measured through a survey adapted from the AIDS Clinical Research Trials Group tool used extensively throughout Kenya and in the Harambee study<sup>13</sup>. Patient activation will be measured through the Patient Activation Measure assessment developed by Insignia Health. Fidelity will be measured as quantity and quality of intervention delivery as intended, comprised of three components: confirmed medication delivery documented by patient e-signature, peer completion of the HIT form, and quality of data entry into the HIT form, which will be assessed by checking for completeness, accuracy and coherent filling of the responses. Completeness of delivery will include these metrics of fidelity in addition to other quality assurance measures centering on medication packaging as well which will be done by the research assistant as the study goes on. We will also conduct surveys with patients, clinicians, and peer delivery agents, focusing on contextual issues impacting implementation, suggestions for modifications, and concepts of feasibility, that is, if the process of delivery and counseling has been successful or not successful in all the settings and the perceived ease of implementing the intervention. We will also evaluate the impact of the pilot on absolute mean change in SBP and medication adherence. The primary adherence outcome is the pill count adherence ratio, which is the proportion of prescribed doses taken over a 1-month time period, assessed at the end of the pilot.

# **Design Team Meeting #6: Iteration II**

#### Session A:

- DT members will engage in icebreaker activities and review previous discussions
- PT4A research team will present and discuss findings from pilot study
- DT will group issues raised in FGDs and from study investigators into themes and propose intervention updates

PT4A Protocol 1.4 23<sup>rd</sup> November, 2022

# Session B:

- DT will create a final intervention model and submit this to the study investigators, research team, and Informatics team
- The research team will conduct individual surveys with DT members to evaluate their experience during the HCD process

The research team and Informatics team will be responsible for creating the final intervention model that will be used for more widespread implementation.

# References

- 1. Chow CK, Teo KK, Rangarajan S, et al. Prevalence, awareness, treatment, and control of hypertension in rural and urban communities in high-, middle-, and low-income countries. JAMA 2013;310:959-68.
- 2. Irazola VE, Gutierrez L, Bloomfield G, et al. Hypertension Prevalence, Awareness, Treatment, and Control in Selected LMIC Communities: Results From the NHLBI/UHG Network of Centers of Excellence for Chronic Diseases. Global Heart 2016;11:47-59.
- 3. Mills KT, Bundy JD, Kelly TN, et al. Global Disparities of Hypertension Prevalence and Control: A Systematic Analysis of Population-Based Studies From 90 Countries. Circulation 2016;134:441-50.
- 4. Whelton PK. The elusiveness of population-wide high blood pressure control. Annual review of public health 2015;36:109-30.
- 5. Roebuck MC, Liberman JN, Gemmill-Toyama M, Brennan TA. Medication adherence leads to lower health care use and costs despite increased drug spending. Health Affairs (Project Hope) 2011;30:91-9.
- Vedanthan R, Kamano JH, Lee H, Andama B, Bloomfield GS, DeLong AK, Edelman D, Finkelstein EA, Hogan JW, Horowitz CR, Manyara S, Menya D, Naanyu V, Pastakia SD, Valente TW, Wanyonyi CC, Fuster V. Bridging Income Generation with Group Integrated Care for cardiovascular risk reduction: Rationale and design of the BIGPIC study. Am Heart J. 2017 Jun;188:175-185. doi: 10.1016/j.ahj.2017.03.012. Epub 2017 Mar 23. PMID: 28577673; PMCID: PMC5491075.
- 7. Aifah A, Okeke NL, Rentrope CR, Schexnayder J, Bloomfield GS, Bosworth H, et al. Use of a human-centered design approach to adapt a nurse-led cardiovascular disease prevention intervention in HIV clinics. Prog Cardiovasc Dis. 2020;63(2):92–100. 18.
- 8. Leung CL, Naert M, Andama B, Dong R, Edelman D, Horowitz C, et al. Human-centered design as a guide to intervention planning for noncommunicable diseases: the BIGPIC study from Western Kenya. BMC Health Serv Res. 2020;20(1):415
- 9. Pittsburgh, PA: linnovating for people: Handbook of human-centered design methods. (2012). LUMA Institute, LLC.
- 10. Parsell G, Gibbs T, Bligh J. Three visual techniques to enhance interprofessional learning. Postgrad Med J 1998;74:387-90.
- 11. Parsell G, Spalding R, Bligh J. Shared goals, shared learning: evaluation of a multiprofessional course for undergraduate students. Med Educ 1998;32:304-11.
- 12. Stuttaford M, Bryanston C, Hundt GL, Connor M, Thorogood M, Tollman S. Use of applied theatre in health research dissemination and data validation: a pilot study from South Africa. Health (London, England: 1997) 2006;10:31-45.
- 13. Odeny TA, et al. Integration of HIV Care with Primary Health Care Services: Effect on Patient Satisfaction and Stigma in Rural Kenya. *AIDS Research and Treatment*. 2013;2013:1-10. doi:10.1155/2013/485715



# **APPENDIX B. STUDY INTERVIEW QUESTIONNAIRES**

Peers and Technology for Adherence, Access, Accountability, and Analytics (PT4A) Study

Study Instrument: Acceptability of Intervention Measure (AIM) for Patients Living with Hypertension

| Study ID: | Date: |
|---|---|
| Age: | Gender: |
| 1. Education/ Elimu | □ No formal education/ Hakuna elimu rasmi |
| □Primary/ Shule ya Msingi | ∃Secondary/ Shule ya Upili |
| □Beyond secondary/ Zaidi ya Shule ya Upili | □Special training e.g Trade. Insert Mafunzo |
| maalum | kwa mfano biashara |
| 2. What is your main source of income?/ Chanz | o chako kikuu cha mapato ni nini? |
| 1 | ss/Trade/Biashara □Teacher/ |
| Uwaalimu | |
| □Health worker/ Mfanyakazi wa afya □Other/s (In | |
| 3. What is your estimated monthly income in Klyanakadiriwa ngapi □KES? <1,000 □1,000 | |
| 9,999 $\square$ >10,000 | 0-2,999 □3,000-4,999 □5,000- |
| 9,999 | |
| 4. How long have you been living with hyperter | nsion/pressure in months? Umeishi kwa |
| muda gani na shinikizo la damu / shinikizo (kwa | a miezi) |
| □<6 months/ Miezi sita □Between 6 months – 1yea | ar/ Kati ya miezi sita na mwaka |
| │<br>│□Between 1-2 years/ Kati ya mwaka mmoja na mb | ili?□>2 years/ Zaidi ya miaka mbili? |
| 5. Where do you mainly seek treatment for hype | |
| babu ya shinikizo la damu | |
| 1 | armacy (over the counter medication) Duka la |
| dawa<br>□Herbalist / Mtaalam wa mimea | (iuu va dawa va kaunta) |
| □Not yet sought care/ Bado sijatafuta huduma □C | (juu ya dawa ya kaunta)<br>Other specify/ Nyingine taja |
| 6. About how long would it take to get from you | |
| you walked to them? Je! Itachukua muda gani l | |
| la dawa lilokaribu ukitembea? | <b>,</b> |
| □Less than 15 minutes/ Chini ya dakika 15 | □16-30 minutes/ Dakika 16-30 |
| □31 minutes to an hour/ dakika 31 hadi saa moja | |
| 7. About how long would it take to get from you walked to them?/ lol tachukus muda gani ki | • |
| you walked to them?/ Je! Itachukua muda gani ku<br>huduma ya afya kilicho karibu ikiwa utatembea kue | |
| Less than 15 minutes/ Chini ya dakika 15 | □16-30 minutes/ Dakika 16-30 |

| ∃31 minutes to an hour/ dakika 31 hadi saa mo | a □More than one hour/ Zaidi ya saa | moia |
|---|---|---|
| Jo i minutes to an nour dakika o i nadi saa mo | a ⊟iviore trian one nour Zaidi ya saa | т тюја |

**Instructions to Study Personnel**: Read all questions aloud to the patient and record answers on questionnaire form.

You were selected to take part in this survey because we value the knowledge you have on our topic of discussion. I kindly request for your honest opinions and ideas. There is no wrong or right response. You should feel free to say whatever you think and feel.

There is a plan to start a project that will support people living with hypertension/pressure at the community level. The purpose of the project is to assist these individuals take hypertension/pressure medication their as required through a peer-led project. A peer will be someone who is living with hypertension/pressure in the community and has been successful in managing their hypertension. The peer will be responsible for a number of things:

- Deliver hypertension medication to people living with hypertension/pressure at their most convenient location (door-to-door medication delivery).
- Provide psychological support to people living with hypertension/pressure during medication delivery and whenever needed.
- Record the health progress of people living with hypertension/pressure in a mobile device whenever they are in contact with a person living with hypertension/pressure.
- Using the mobile device, communicate with a clinician where the individuals living with hypertension receive care to discuss their health progress.
- Whenever necessary enable a conversation (either audio or video) between the clinician and the patient using the mobile device at the patient's convenient location.
- Insert the revised prototype

| | Completely disagree | Disa-<br>gree | Neither<br>agree nor<br>disagree | Agree | Complet<br>agree |
|---|---|---|---|---|---|
| The HIT-Peer Delivery system meets my needs | ① | 2 | 3 | 4 | (5) |
| 2. The HIT-Peer Delivery system is appealing to me. | ① | 2 | 3 | 4 | (5) |
| 3. I like the HIT-Peer Delivery system. | 0 | 2 | 3 | 4 | (5) |
| 4. I would like to be enrolled in the HIT-Peer Delivery system. | ① | 2 | 3 | 4 | (5) |

With this revisions to our PT4A strategy, will this prototype do the following for you.

# Intervention Appropriateness Measure (IAM)

| | Completely disagree | Disa-<br>gree | Neither<br>agree<br>nor dis-<br>agree | Agree | Comple<br>agree |
|---|---|---|---|---|---|
| he HIT-Peer Delivery system seems fitting. | 1 | 2 | 3 | 4 | (5) |
| he HIT-Peer Delivery system seems suita- | ① | 2 | 3 | 4 | (5) |
| he HIT-Peer Delivery system seems applile. | ① | 2 | 3 | 4 | (5) |
| he HIT-Peer Delivery system seems like a d match. | ① | 2 | 3 | 4 | (5) |

Total Score:

# Peers and Technology for Adherence, Access, Accountability, and Analytics (PT4A) Study

Study Instrument: Acceptability of Intervention Measure (AIM) for Health Care Team

| Study ID: | Date: | | | |
|---|---|---|---|---|
| Age: | Gender: | | | |
| 1. What is your primary role at the facility? | <br> | | | |
| □MO □CO □Nurse □Other staff (specify) | | | | |
| 2. How long have you served as a health prov | rider for Hypert | ensive patie | ents? | |
| 3. What is your interaction with patients living | with Hypertens | sion? | | |
| Instructions to Study Personnel: Read all q answers on questionnaire form. | uestions aloud | to the healt | thcare provide | er and record |
| You were selected to take part in this survey to topic of discussion. I kindly request for your heresponse. You should feel free to say whatever there is a plan to start a project that will suppose community level. The purpose of the project is sure medication their as required through a pewith hypertension/pressure in the community at tension. The peer will be responsible for a nure. Deliver hypertension medication to perconvenient location (door-to-door med). Provide psychological support to peoption delivery and whenever needed. Record the health progress of people is whenever they are in contact with a pewing the mobile device, communicated pertension receive care to discuss their whenever necessary enable a conversand the patient using the mobile device. Insert the revised prototype | onest opinions or you think an ort people living to assist these eer-led project. and has been some of things: ople living with hydrony with hydrony with a clinicial ir health progresation (either a sation (either a serious property of the serious of the seriou | and ideas. Id feel. g with hyper e individuals A peer will is hypertension/ ertension/pre in hypertensi n where the ess. eudio or vide | There is no writension/press take hyperte be someone with managing the on/pressure at the someone with the source in a motion/pressure in a motion/pressure in a motion/pressure in dividuals live to between the source of the source in the source of the source in the source in the source in the source of the source in the source is not the source in th | rong or right sure at the ension/pres- who is living neir hyper- their most ng medica- pobile device ving with hy- |
| | Completely | Dieggroo | Neither | Agree C |
| | disagree | Disagree | agree nor<br>disagree | Agree |

| The HIT-Peer Delivery system meets the patients needs | ① | 2 | 3 | 4 |
|---|---|---|---|---|
| 2. The HIT-Peer Delivery system is appealing to both the patient and I healthcare provider | ① | 2 | 3 | 4 |
| 3. I like the HIT-Peer Delivery system. | 1 | 2 | 3 | 4 |
| 4. I would like my patients enrolled in the HIT-Peer Delivery system. | ① | 2 | 3 | 4 |

# With this revisions to our PT4A strategy, will this prototype do the following for you.

# **Intervention Appropriateness Measure (IAM)**

| | Completely disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Completely agree |
|---|---|---|---|---|---|
| The HIT-Peer Delivery system seems fitting. | ① | 2 | 3 | 4 | (5) |
| 2. The HIT-Peer Delivery system seems suitable. | ① | 2 | 3 | 4 | (5) |
| 3. The HIT-Peer Delivery system seems applicable. | ① | 2 | 3 | 4 | (5) |
| 4. The HIT-Peer Delivery system seems like a good match. | ① | 2 | 3 | 4 | (5) |

Weiner, B.J., Lewis, C.C., Stanick, C. *et al.* Psychometric assessment of three newly developed implementation outcome measures. *Implementation Sci* **12**, 108 (2017). https://doi.org/10.1186/s13012-017-0635-3

# Peers and Technology for Adherence, Access, Accountability, and Analytics (PT4A) Study

Study Instrument: Acceptability of Intervention Measure (AIM) for PEERS

| Study ID: | Date: |
|---|---|
| Age: | Gender: |
| 1. Education/ Elimu | No formal education/ Hakuna elimu rasmi |
| □Primary/ Shule ya Msingi □Se | condary/ Shule ya Upili |
| □Beyond secondary/ Zaidi ya Shule ya Upili □<br>maalum | Special training e.g Trade. Insert Mafunzo |
| | kwa mfano biashara |
| | rade/Biashara |
| ☐ Health worker/ Mfanyakazi wa afya ☐ Other/s (Insert | :): Ingine |
| 3. How long have you worked as a peer? | |
| 4. What is your estimated monthly income in KES? | <sup>2</sup> / Je! Mapato yako ya kila mwezi yanakadiriwa |
| ngapi □KES?<1,000 □1,000-2,999 □3,000-4,99 | 99 □5,000-9,999 □>10,000 |
| 5. How long have you been living with hypertensio | n/pressure in months? Umeishi kwa muda |
| gani na shinikizo la damu / shinikizo (kwa miezi) <6 months/ Miezi sita Between 6 months – 1year/ k | Kati va miezi sita na mwaka |
| · | • |
| □Between 1-2 years/ Kati ya mwaka mmoja na mbili?□ | |
| 6. Where do you mainly seek treatment for hyperte shinikizo la damu | nsion/pressure?/ Unapata wapi matibabu ya |
| | acy (over the counter medication) Duka la dawa |
| □Herbalist / Mtaalam wa mimea | (juu ya dawa ya kaunta) |
| □Not yet sought care/ Bado sijatafuta huduma □Othe | |
| 7. About how long would it take to get from your he walked to them? Je! Itachukua muda gani kutoka n | |
| lokaribu ukitembea? | □16-30 minutes/ Dakika 16-30 |
| □Less than 15 minutes/ Chini ya dakika 15 | 10-30 Illillutes/ Dakika 10-30 |
| □31 minutes to an hour/ dakika 31 hadi saa moja | □More than one hour/ Zaidi ya saa moja |
| 8. About how long would it take to get from your he | |
| walked to them?/ Je! Itachukua muda gani kutoka nyi | umbani kwako kwenda kituo cha huduma ya afya |
| kilicho karibu ikiwa utatembea kuelekea huko?<br>□Less than 15 minutes/ Chini ya dakika 15 | □16-30 minutes/ Dakika 16-30 |
| □31 minutes to an hour/ dakika 31 hadi saa moja | □More than one hour/ Zaidi ya saa moja |

**Instructions to Study Personnel:** Read all questions aloud to the patient and record answers on questionnaire form.

You were selected to take part in this survey because we value the knowledge you have on our topic of discussion. I kindly request for your honest opinions and ideas. There is no wrong or right response. You should feel free to say whatever you think and feel.

There is a plan to start a project that will support people living with hypertension/pressure at the community level. The purpose of the project is to assist these individuals take hypertension/pressure medication their as required through a peer-led project. A peer will be someone who is living with hypertension/pressure in the community and has been successful in managing their hypertension. The peer will be responsible for a number of things:

- Deliver hypertension medication to people living with hypertension/pressure at their most convenient location (door-to-door medication delivery).
- Provide psychological support to people living with hypertension/pressure during medication delivery and whenever needed.
- Record the health progress of people living with hypertension/pressure in a mobile device whenever they are in contact with a person living with hypertension/pressure.
- Using the mobile device, communicate with a clinician where the individuals living with hypertension receive care to discuss their health progress.
- Whenever necessary enable a conversation (either audio or video) between the clinician and the patient using the mobile device at the patient's convenient location.
- Insert the revised prototype

| | Γ | <b>.</b> | T | T | 1 |
|---|---|---|---|---|---|
| | Completely disa-<br>gree | Disagree | Neither<br>agree nor<br>disagree | Agree | Comple<br>agree |
| The HIT-Peer Delivery system meets my needs | ① | 2 | 3 | 4 | (5) |
| 2. The HIT-Peer Delivery system is appealing to me. | ① | 2 | 3 | 4 | \$ |
| 3. I like the HIT-Peer Delivery system. | ① | 2 | 3 | 4 | (5) |
| 4. I would like to be enrolled in the HIT-Peer Delivery system. | ① | 2 | 3 | 4 | (5) |

With this revisions to our PT4A strategy, will this prototype do the following for you?

# **Intervention Appropriateness Measure (IAM)**

| | Completely disagree | Disagree | Neither<br>agree<br>nor dis-<br>agree | Agree | Complete<br>agree |
|---|---|---|---|---|---|
| The HIT-Peer Delivery system seems fitting. | 1 | 2 | 3 | 4 | (5) |
| The HIT-Peer Delivery system seems suitable. | 1) | 2 | 3 | 4 | (5) |
| The HIT-Peer Delivery system seems applicae. | ① | 2 | 3 | 4 | (5) |
| The HIT-Peer Delivery system seems like a pod match. | 1 | 2 | 3 | 4 | (5) |

Total Score:

# Subaim 2.2: Conduct a pilot of the intervention and evaluate feasibility

# AIM 2.2 Study Instrument: EVALUATION OF FEASIBILITY QUESTIONNAIRE FOR PATIENTS

| Hello, my name is I am a research assistant for the PT4A study. I am approaching you as you have participated as a patient in the PT4A program and as such our feedback would be helpful for the program. I would like to ask you some questions to learn about your experiences with the PT4A program. I will ask you questions about your physical health, your mental health, and how you feel when you interact with a peer from the PT4A program. Your answers will help me understand what types of services people who are living with high blood pressure need to stay healthy. |
|---|
| Do you have any questions? |
| Ok, let's begin |
| Now I would like to hear about your experience with the PT4A peer delivery program. Please answer honestly and to the best of your knowledge. All responses are confidential. |
| 1. When you receive medication and counseling from a peer, how often do the peers treat you with courtesy and respect? All the time Some of the time None of the time |
| 2. When you receive medication and counseling from a peer, how often do the peers listen carefully to you? All the time A lot of the time Some of the time None of the time |
| <ul> <li>3. When you receive medication and counseling from a peer, how often do the peers ask for your opinion regarding your healthcare?</li> <li>All the time</li> <li>A lot of the time</li> <li>Some of the time</li> <li>None of the time</li> </ul> |
| <ul> <li>4.When you receive medication and counseling from a peer, how often are you satisfied with the amount of time your peer spends with you?</li> <li>All the time</li> <li>A lot of the time</li> <li>Some of the time</li> <li>None of the time</li> </ul> |

| Please tell me how much you agree or disagree with the following statements |
|---|
| 5. The peers in the PT4A delivery program can be trusted to keep my medical information private and |
| confidential. |
| □ Strongly agree |
| □ Agree |
| □ Disagree |
| □ Strongly Disagree |
| 6.Whenever you had questions about your medications or health which you brought up to the peer, |
| how often were you satisfied about the answers you received from the peer? |
| ☐ All the time |
| □ A lot of the time |
| □ Some of the time |
| □ None of the time |
| 7. When you receive medication and counseling from a peer, how often did you get clear instructions |
| on how to use/take the medication? |
| ☐ All the time |
| □ A lot of the time |
| □ Some of the time |
| □ None of the time |
| 8. Did you feel the peer having the Mobile Device helped with record keeping for the next clinical en- |
| counter you had with your doctor? |
| □ Strongly agree |
| ☐ Agree |
| □ Disagree |
| □ Strongly Disagree |
| 9. Did the Mobile Device help you have a consultation with a healthcare provider for any emerging |
| medical issue? Yes No |
| Do you feel that the use of the mobile device helped you to manage the arising medical issue that |
| came up? |
| □ Strongly agree |
| ☐ Agree |
| ☐ Disagree |
| □ Strongly Disagree |
| 10. Did the use of a peer to deliver medication has improve your health? |
| □ Strongly agree |
| ☐ Agree |
| □ Disagree |
| □ Strongly Disagree |
| 11. Did the use of a peer to offer psychosocial support help you improve your quality of life? |
| □ Strongly agree |
| □ Agree |
| □ Disagree |

| Strongly Disagree | |
|---|---|
| 11. Has the use of a peer to deliver medication helped you to adhere to medication and you hav | e expe- |
| rienced few if no symptoms associated with Hypertension | |
| □ Strongly agree | |
| □ Agree | |
| □ Disagree | |
| Strongly Disagree | |
| AIM 2.2 Study Instrument: EVALUATION OF DELIVERY PROCESS AND COMPLETENESS | |
| QUESTIONNAIRE FOR PATIENTS | |
| Now I would like to hear about your feedback on the PT4A medication delivery process. | |
| Please answer honestly and to the best of your knowledge. All responses are confidential. | |
| Successful/proper deliveries | |
| The peers delivered the right medication as requested | |
| ☐ All the time | |
| □ A lot of the time | |
| □ Some of the time | |
| □ None of the time | |
| The medication was delivered on the date expected | |
| ☐ All the time | |
| □ A lot of the time | |
| □ Some of the time | |
| □ None of the time | |
| The medication was delivered at the time expected | |
| ☐ All the time | |
| □ A lot of the time | |
| □ Some of the time | |
| □ None of the time | |
| Medication packaging | |
| The medication was properly sealed during the delivery | |
| □ All the time | |
| □ A lot of the time | |
| □ Some of the time | |
| □ None of the time | |
| The medication was properly labeled and the dosage indicated | |
| □ All the time | |
| □ A lot of the time | |
| □ Some of the time | |
| □ None of the time | |
| The medication was properly labeled and the dosage indicated | |
| □ All the time | |
| □ A lot of the time | |
| □ Some of the time | |
| □ None of the time | |
| The peer was able to give you instructions for medication use | |
| ☐ All the time | |

PT4A Protocol 1.4 23<sup>rd</sup> November, 2022

| □ A lot of the time |
|---------------------------------------------------------------------|
| □ Some of the time |
| □ None of the time |
| The medication brand changes were clearly communicated |
| □ All the time |
| □ A lot of the time |
| □ Some of the time |
| □ None of the time |
| The medication payments reflected the amount of medication received |
| □ All the time |
| □ A lot of the time |
| □ Some of the time |
| □ None of the time |
| Total Scores |

#### APPENDIX C. INTERVIEW GUIDES FOR FEASIBILITY EVALUATION

# Peers and Technology for Adherence, Access, Accountability, and Analytics (PT4A) Study

Study Instrument: Focus Group Discussion (FGD) Guide for Clinical Team

| FGD moderator: | <br><del>_</del> |
|-----------------|------------------|
| FGD note taker: | <br> |
| Date://2022 | |
| County: | |
| Start Time: | |
| End Time: | |

#### FGD:

- Inform the participants about the study guided by the study information sheet.
- Provide participants with an opportunity to ask questions.
- Obtain written consent from each participant privately. (2 copies per participants)
- Provide each participant with a copy of their signed informed consent form.
- Complete the demographic survey for each participant privately.

# **Demographic Survey**

| Indicate or insert your res | sponses as n | ecessary | | | |
|---|---|---|---|---|---|
| 1. Study ID: | | | | | |
| 2. State your age (Years) | | | | | |
| 3. Sex | Male | Female | | | |
| 4. What is your primary role at the facility? | МО | CO | Nurse | | Other staff (specify) |
| 5. How long have you served as a health provider? | | | | | |
| 6. Have you interacted with patients living with Hypertension? | Yes | | 1 | No | |

NB: To be completed for each participant

| | Summary of observations during FGD | |
|---|---|---|
| <u>Mo</u><br>sic | oderator and note taker: In the space below, please provide a summary of on you just had including both verbal and nob-verbal cues. | the FGD ses- |
| PT | 4A Protocol 1.4 23 <sup>rd</sup> November, 2022 | Page <b>61</b> of <b>9</b> 6 |
| | | Page <b>61</b> of <b>86</b> |

# Focus Group Discussion Guide Clinical Team

| ************ | ***** |
|---|---|
| for welcoming us to your community. notes during our discussions. We will also the participants the tape recorder). This will anything. Your opinions and experiences are | and I will help guide our discussion today. Thank you XXX is also present today to help take be recording this session using a tape recorder (show help us capture what you say without missing out on re very important to us since it will help us understand dividuals living with hypertension in your community. |
| experience in PT4A program I kindly required wrong or right response. You should feel fr | ession because we value your feedback regarding your est for your honest opinions and ideas. There is no ree to say whatever you think and feel. You are welnt. I am eager to hear what you have to say. Do you so far? |

# FGD rules

Before we start, I would like as to you mention some of the rules that will guide our discussion

- 1. There are no right or wrong answers. We expect that you will have differing points of view. Please feel free to share your point of view even if it differs from what others have said.
- We are recording this session as we discussed, because we do not want to miss any of your comments. No names will be included in any reports. Your comments are confidential. Please speak loudly for I want to be accurate in capturing what you say.
- 3. Don't feel like you have to respond all the time. But if you want to follow up on something that someone has said, you want to agree, or disagree, or give an example, feel free to do that.
- 4. I am here to ask questions, listen, and make sure everyone has a chance to share. We're interested in hearing from each of you. So if you are talking a lot, I may ask you to give others a chance. We just want to make sure all of you have a chance to share your ideas.
- 5. If you have a cell phone, please put it on quiet mode.

Now let us start discussions about your perceptions about the PT4A Intervention.

#### A. PT4A intervention:

PT4A project was started to support people living with hypertension/pressure at the community level. The purpose of the project was to assist these individuals take hypertension/pressure medication as required through a peer-led project. This peer led project used a mobile device similar to regular mobile phone, a smart phone, or a tablet. The mobile device enabled us to deliver hypertension health services to the patients in a safe, confidential, and timely manner. The device, supported patients in treatment counseling; delivering medications to the patients; accounting for the types of medications delivered, quantity, and amount of fees the patients pays at the time of delivery (like an Mpesa transaction); and also connecting the patients with their doctor whenever they needed.. In doing so, a peer collected health information from the patients on a regular basis on this mobile device.

A peer was someone living with hypertension/pressure in the community who had been successful in managing their hypertension. The peer was responsible for a number of things:

- Delivering hypertension medication to people living with hypertension/pressure at their most convenient location (door-to-door medication delivery).
- Confirming payment of medication (Mpesa transaction) by people living with hypertension/pressure before issuing the medication.
- Providing psychological support to people living with hypertension/pressure during medication delivery and whenever needed.
- Recording the health progress of people living with hypertension/pressure in a mobile device whenever they are in contact with a person living with hypertension/pressure.
- Using the mobile device, communicate with a clinician, to discuss the progress of an individual living with hypertension.
- Whenever it was necessary, they enabled a conversation (<u>intervention</u>: either audio or video) between the clinician and the patient using the mobile device at the patient's convenient location.
- 1. What did you think about this peer-led project in supporting individuals living with hypertension in the community?

### Probe:

- What parts of the project did you like? Why?
- What part of the project didn't you like? Why?
- Parts of the project that were easily carried out? Why?
- Parts of the project that were difficult to carry out? Why?
- 2. What were the advantages of this kind of peer-led program? Probe:
  - Advantages of peers leading the delivery of health services
  - Advantages of door to door drug delivery
  - Advantages of peers providing psychological support to individuals living with hypertension at the community level
  - Advantages of peers recording health information of the individuals receiving hypertension medication at the community on the mobile device (Probe: quality of care, provider-patient communication, privacy and confidentiality)

- Advantages of doctor and the patient having a clinical meeting using a mobile device at the community level (Probe: quality of care, provider-patient communication, privacy and confidentiality)
- 3. What were the disadvantages of this kind of peer-led program? Probe:
  - Disadvantages of peers leading the delivery of health services
  - Disadvantages of door to door drug delivery
  - Disadvantages of peers providing psychological support to individuals living with hypertension at the community level
  - Disadvantages of peers recording health information of the individuals receiving hypertension medication at the community on the mobile device (Probe: quality of care, provider-patient communication, privacy and confidentiality)
  - Disadvantages of doctor and the patient having a clinical meeting using a mobile device at the community level (Probe: quality of care, provider-patient communication, privacy and confidentiality)
- 4. In what ways did this peer-led program affect the management of hypertension at the community level?

Probe:

- How did it affect medication adherence for individuals living with hypertension?
- How did it affect follow-up of individuals living with hypertension?
- How did it effect on how hypertension is perceived in the community?
- 5. In what ways did this peer-led program affect the management of hypertension at the facility level?

Probe:

- Positive effects (How did this program complement the efforts in clinic?)
- Negative effects (How did this make it challenging to manage hypertension at the clinic level
- 6. In what ways did this peer-led affect the way care for hypertension/pressure is offered during the current COVID pandemic?
  - B. Peers

Now let us talk more specifically about the peers who delivered these health services to individuals living with hypertension at the community.

7. What are your perception about the peers that were used to implement the PT4A intervention

Probe:

- characteristics of the peer
- Qualifications/skill
- Training
- Integrity
- C. Mobile device

Now let us talk more about the mobile device used to deliver these health services to individuals living with hypertension at the community.

- 8. What is your perception of mobile device used by the peers to deliver the PT4A intervention?
- 9. What are the mobile device features that were most useful in implementing the PT4A intervention?

#### Probe:

- Type of device
- Size of device
- Connectivity
- Content
- Data flow
- Care facilitation features
- 10. What were the mobile device features that were not useful in implementing the PT4A intervention?

#### Probe:

- Type of device
- Size of device
- Connectivity
- Content
- Data flow
- Care facilitation features
- 11. What was your perception about the mobile payment mode used to pay for the Hypertension medications in the PT4A intervention?
- 12. How did the use of a mobile device impact the delivery of hypertension services at the community?
  - D. Recommendation for improving the PT4A project

We are about to end our discussion today. But before we end, we would like to hear about some of your recommendations for improving the proposed peer-led project to support individuals living with hypertension.

- 13. What is your perception about the uptake of this peer led project in your facility?
- 14. Would you recommend this peer-led project to other individuals living with HTN? Why
- 15. What would be your recommendation for improving this peer-led project? Probe:
  - Parts of the project that could be improved. How?
- 16. What would make this peer led project acceptable as part of standard care?
- 17. What would make this peer-led project sustainable?

### E. Closing

We have now come to the end of our discussions today. Thank you for your time and participation. We very much appreciate your comments, discussion, and input. We plan to take into account everything that was said today as we continue to improve the services we offer to your community.

Do you have any questions related to our discussion today?

#### NB: Before ending

- Remind participants about the confidentiality of the interview.
- Ask if there is anything that wasn't raised that should have been that is important to know in understanding their perception about the peer-led intervention.
- Offer lunch stipend and provide contact information for any future questions they may have.
- Thank participants once again for their time.

Peers and Technology for Adherence, Access, Accountability, and Analytics (PT4A) Study/

Study Instrument: Focus Group Discussion (FGD) Guide for Individuals living with Hypertension

| FGD moderator/ Msimamizi: |
|---|
| FGD note taker/ Mchukua noti: |
| Date/ Tarehe://2022 |
| County/ Kaunti: |
| Category of FGD (tick)/ Aina ya Majadiliano ya Kikundi [] Men living with hypertension / Wanaume wanoishi na Shinikizo la damu/ Pressure [] Women living with hypertension/ Wanawake Wanaoishi na Shinikizo la damu/ Pressure sure []Community members/ Wanachama wa Jamii |
| Start Time/ Saa ya Kuanza: |
| End Time/ Saa ya Kumaliza: |

#### FGD:

- Inform the participants about the study guided by the study information sheet.
- Provide participants with an opportunity to ask questions.
- Obtain written consent from each participant privately. (2 copies per participants)
- Provide each participant with a copy of their signed informed consent form.
- Complete the demographic survey for each participant privately.

# **Demographic Survey for Individuals Living with Hypertension**

| Indicate or insert your re | sponses as ne | cessary | | | |
|---|---|---|---|---|---|
| 1. Study ID:/ Nambari ya | Utafiti: | | | | |
| 2. State your age (Year of Birth)/ <i>Taja umri wako</i> ( <i>Mwaka wa kuzaliwa</i> ) | | | | | |
| 3. Sex/ <i>Jinsia</i> | □Male<br><i>Kiume</i> ) | □Female <i>(K</i> | ike) | | |
| 4. Education/ <i>Elimu</i> | □No formal<br>education/<br><i>Hakuna</i><br><i>elimu rasmi</i> | □Primary/<br>Shule ya<br>Msingi | □Second-<br>ary/ <b>Shule</b><br><b>ya Upili</b> | □Beyond<br>second-<br>ary/<br>Zaidi ya<br>Shule ya<br>Upili | □Special training e.g<br>Trade. <i>Insert</i><br><i>Mafunzo maalum</i><br><i>kwa mfano biashara</i> |
| 5. What is your main source of income?/ Chanzo chako kikuu cha mapato ni nini? | □Farming/<br><i>Ukulima</i> | □Busi-<br>ness/<br>Trade/ <b>Bi-</b><br>ashara | □Teacher/<br><b>Uwaalimu</b> | □Health<br>worker/<br><i>Mfanyak</i><br><i>azi wa</i><br><i>afya</i> | □Other/s (Insert): In-<br>gine |
| 6. What is your estimated monthly income in KES?/ Je! Mapato yako ya kila mwezi yanakadiriwa pesa ngapi (Kes? | □<1,000 | □1,000-<br>2,999 | □ 3,000-<br>4,999 | □ 5,000-<br>9,999 | □ >10,000 |
| 8. How long have you been living with hypertension/pressure in months? Umeishi na shinikizo la damu / pressure (kwa miezi ngapi | □<6 months/<br><i>Miezi sita</i> | □Between 6 months –<br>1year/ <i>Kati ya miezi</i><br><i>sita na mwaka?</i> | | □Be- tween 1- 2 years Kati ya mwaka mmoja na mbili? | □>2 years/ <b>Zaidi ya</b><br>miaka mbili? |
| 9. Where do you mainly seek treatment for hypertension/pressure? / Unapata wapi matibabu ya shinikizo la damu/ pressure | □Health facility/ <i>Kituo</i> cha afya/ name the health facility | □Phar- macy (over the counter medica- tion) <i>Duka la dawa / dawa ya kaunta</i> ) | □Herbalist<br>/ Mtaalam<br>wa dawa<br>za<br>Kienyeji | □Not yet sought care/ Bado sijatafut a huduma | □Other specify/ <i>Nyingine taja</i> |

| 10. About how long would it take to get from your home to the nearest chemist/pharmacy if you walked to them? <i>Je!</i> Itachukua muda gani kutoka nyumbani kwako kwenda kwa duka la dawa lilokaribu ukitembea? | □Less than<br>15 minutes/<br>Chini ya<br>dakika 15 | □16-30<br>minutes/<br><i>Dakika</i><br>16-30 | □31 minutes to an hour/ dakika 31 hadi saa moja | □More than one hour/ <b>Zaidi ya</b> saa moja |
|---|---|---|---|---|
| 11. About how long would it take to get from your home to the nearest healthcare facility if you walked to them?/Je! Itachukua muda gani kutoka nyumbani kwako kwenda kituo cha huduma ya afya kilicho karibu ikiwa utatembea kuelekea huko? | □Less than<br>15 minutes/<br>Chini ya<br>dakika 15 | □16-30<br>minutes/<br><i>Dakika</i><br>16-30 | □31 minutes to an hour/ dakika 31 hadi saa moja | □More than one hour/ <b>Zaidi ya</b> saa moja |

NB: To be completed for each participant

| Summary of observations during FGD | |
|---|---|
| Moderator and note taker: In the space below, please provide a su sion you just had including both verbal and nob-verb | ummary of the FGD ses-<br>pal cues. |
| PT4A_Peer team Interview Guide Post-Intervention. | Page <b>70</b> of <b>86</b> |

# <u>Focus Group Discussion Guide</u> Individuals living with Hypertension

| ******** | ****** | ****** | ***** | **** | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Opening Re | <u>emarks</u> | | | | | | | | | |
| Hello. M | ly name | is | _XXX | _ and I | will | help | guide | our di | iscussio | n today |
| XXX | | _ is also | present today to | o help ta | ake no | otes d | uring o | ur disc | cussions | . We will |
| also be rec | ording thi | s session | i using a tape re | ecorder ( | (show | the p | articipa | ants th | e tape r | ecorder). |
| This will he | lp us capt | ure what | you say without | missing | out or | n any | thing. Y | our op | oinions a | ind expe- |
| riences are | very imp | ortant to ι | us since it will h | elp us ur | nderst | and h | ow to | develo | p health | program |
| to assist me | ore people | e living wit | th hypertension | in your c | ommı | unity. | | | | |
| You were s | selected to | take par | t in this discuss | ion beca | use v | ou pa | rticipat | ed in t | his stud | v and we |

You were selected to take part in this discussion because you participated in this study and we value your experiences and knowledge on our topic of discussion. I kindly request for your honest opinions and ideas. There is no wrong or right response. You should feel free to say whatever you think and feel. You are welcome to say as much or as little as you want. I am eager to hear what you have to say. Do you have any questions about what I have said so far?

### FGD rules

Before we start, I would like as to you mention some of the rules that will guide our discussion

- 6. There are no right or wrong answers. We expect that you will have differing points of view. Please feel free to share your point of view even if it differs from what others have said.
- 7. We are recording this session as we discussed, because we do not want to miss any of your comments. No names will be included in any reports. Your comments are confidential. Please speak loudly for I want to be accurate in capturing what you say.
- 8. Don't feel like you have to respond all the time. But if you want to follow up on something that someone has said, you want to agree, or disagree, or give an example, feel free to do that.
- 9. I am here to ask questions, listen, and make sure everyone has a chance to share. We're interested in hearing from each of you. So if you are talking a lot, I may ask you to give others a chance. We just want to make sure all of you have a chance to share your ideas.
- 10. If you have a cell phone, please put it on quiet mode.
### A. PT4A intervention:

PT4A project was started to support people living with hypertension/pressure at the community level. The purpose of the project was to assist these individuals take hypertension/pressure medication as required through a peer-led project. This peer led project used a mobile device similar to regular mobile phone, a smart phone, or a tablet. The mobile device enabled us to deliver hypertension health services to the patients in a safe, confidential, and timely manner. The device, supported patients in treatment counseling; delivering medications to the patients; accounting for the types of medications delivered, quantity, and amount of fees the patients pays at the time of delivery (like an Mpesa transaction); and also connecting the patients with their doctor whenever they needed.. In doing so, a peer collected health information from the patients on a regular basis on this mobile device.

A peer was someone living with hypertension/pressure in the community who had been successful in managing their hypertension. The peer was responsible for a number of things:

- Delivering hypertension medication to people living with hypertension/pressure at their most convenient location (door-to-door medication delivery).
- Confirming payment of medication (Mpesa transaction) by people living with hypertension/pressure before issuing the medication.
- Providing psychological support to people living with hypertension/pressure during medication delivery and whenever needed.
- Recording the health progress of people living with hypertension/pressure in a mobile device whenever they are in contact with a person living with hypertension/pressure.
- Using the mobile device, communicate with a clinician, to discuss the progress of an individual living with hypertension.
- Whenever it was necessary, they enabled a conversation (<u>intervention</u>: either audio or video) between the clinician and the patient using the mobile device at the patient's convenient location.

I would first like to ask you questions regarding your perception and experience with the PT4A project

18. What did you think about this peer-led project in supporting you as an individual living with hypertension in the community?

## Probe:

- What parts of the project did you like? Why?
- What part of the project didn't you like? Why?
- 19. What were your experiences with peers leading the delivery of hypertension services in the community?

# Probe:

- What did you like? Why?
- What didn't you like? Why?
- 20. What were your experiences with peers delivering medication at your convenient location in the community?

#### Probe:

- What did you like? Why?
- What didn't you like? Why?

PT4A Peer team Interview Guide Post-Intervention.

21. What were your experiences with peers providing psychological support to you in the community?

Probe:

- What did you like? Why?
- What didn't you like? Why?
- 22. What is your perception of peers recording your health information on a mobile device? Probe:
  - Privacy and confidentiality.
- 23. What is your perception of you and the doctor having a clinical meeting using a mobile device at the community?

Probe:

- Quality of care
- Provider-patient communication
- Privacy and confidentiality
- 24. What is your perception about the mobile payment mode used to pay for the Hypertension medications in the PT4A intervention?
- 25. What are your perceptions about the characteristics of the peers who delivered the hypertension services to your at the community?

Probe:

- Age
- Gender
- Personality
- Academic qualification
- Skill/Training
- 26. In what ways did this peer-led program affect your hypertension care? Probe:
  - How did it affect your medication adherence?
  - How did it affect your clinic adherence?
  - How did it affect the quality of care you received?
  - B. Recommendation for improving the PT4A project

We are about to end our discussion today. But before we end, we would like to hear about some of your recommendations for improving this peer-led project to support individuals living with hypertension/pressure

- 27. Would you recommend this peer-led project to other individuals living with HTN? Why
- 28. What would be your recommendation for improving this peer-led project? Probe:
  - Parts of the project that could be improved. How?
  - C. Closing

We have now come to the end of our discussions today. Thank you for your time and participation. We very much appreciate your comments, discussion, and input. We plan to take into account everything that was said today.

Do you have any questions related to our discussion today?

# NB: Before ending

- Remind participants about the confidentiality of the interview.
- Ask if there is anything that wasn't raised that should have been that is important to know in understanding their perception about the peer-led intervention.
- Offer lunch stipend and provide contact information for any future questions they may have.
- Thank participants once again for their time.

# Peers and Technology for Adherence, Access, Accountability, and Analytics (PT4A) Study

Study Instrument: Key Informant Interview Guide for Peers Team.

| FGD moderator: |
|-----------------|
| FGD note taker: |
| Date:/2022 |
| County: |
| Start Time: |
| End Time: |
| Life Tillie. |

#### FGD:

- Inform the participants about the study guided by the study information sheet.
- Provide participants with an opportunity to ask questions.
- Obtain written consent from each participant privately. (2 copies per participants)
- Provide each participant with a copy of their signed informed consent form.
- Complete the demographic survey for each participant privately.

# **Demographic Survey**

| Indicate or insert your responses as necessary | | |
|---|---|---|
| 1. Study ID: | | |
| 2. State your age (Years) | | |
| 3. Sex | Male | Female |
| 5. How long have you served as a peer? | | |
| 6. How long have you interacted with patients living with Hypertension? | | |

NB: To be completed for each participant

# Key Informant Interview Guide Peers Team

| ********************************** |
|---|
| Opening Remarks |
| Hello. My name isXXX and I will help guide our discussion today. Thank you for welcoming us to your communityXXX is also present today to help take notes during our discussions. We will also be recording this session using a tape recorder (show the participants the tape recorder). This will help us capture what you say without missing out on anything. Your opinions and experiences are very important to us since it will help us understand how helpful the intervention was for patients with hypertension. |
| You were selected to take part in this discussion because we value your feedback regarding your experience in PT4A program. I kindly request for your honest opinions and ideas. There is no wrong or right response. You should feel free to say whatever you think and feel. You are welcome to say as much or as little as you want. I am eager to hear what you have to say. Do you have any questions about what I have said so far? |
| FGD rules |
| Before we start, I would like as to you mention some of the rules that will guide our discussion |
| <ol> <li>There are no right or wrong answers. We expect that you will have differing points of view.</li> <li>Please feel free to share your point of view</li> </ol> |
| <ol> <li>We are recording this session as we discussed, because we do not want to miss any of<br/>your comments. No names will be included in any reports. Your comments are confiden-<br/>tial. Please speak loudly for I want to be accurate in capturing what you say.</li> </ol> |
| 3. I am here to ask questions, listen, and make sure everyone has a chance to share. We're interested in hearing from each of you. So if you are talking a lot, I may ask you to give others a chance. We just want to make sure all of you have a chance to share your ideas. |
| 4. If you have a cell phone, please put it on quiet mode. |

Now let us start our discussion with talking about how the project was perceived and the impact it had on individuals living with hypertension.

#### D. PT4A intervention:

There is a plan to start a project that will support people living with hypertension/pressure at the community level. The purpose of the project is to assist these individuals take hypertension/pressure medication as required through a peer-led project. This peer led project will use a mobile device similar to regular mobile phone, a smart phone, or a tablet. The mobile device will enable us to deliver hypertension health services to the patients in a safe, confidential, and timely manner. With the device, we will support the patients in treatment counseling; delivering medications to the patients; accounting for the types of medications delivered, quantity, and amount of fees the patients pays at the time of delivery (like an Mpesa transaction); and also connecting the patients with their doctor whenever they need. To do so, a peer will need to collect health information from the patients on a regular basis on this mobile device.

A peer will be someone who is living with hypertension/pressure in the community and has been successful in managing their hypertension. The peer will be responsible for a number of things:

- Deliver hypertension medication to people living with hypertension/pressure at their most convenient location (door-to-door medication delivery).
- Confirm payment of medication (Mpesa transaction) by people living with hypertension/pressure before issuing the medication.
- Provide psychological support to people living with hypertension/pressure during medication delivery and whenever needed.
- Record the health progress of people living with hypertension/pressure in a mobile device whenever they are in contact with a person living with hypertension/pressure.
- Using the mobile device, communicate with a clinician, to discuss the progress of an individual living with hypertension.
- Whenever necessary enable a conversation (<u>intervention</u>: either audio or video) between the clinician and the patient using the mobile device at the patient's convenient location.

I would first like to ask you questions regarding your perception and experience with the PT4A project

- 1. Could you kindly describe your role in the PT4A intervention?
- 2. What was your general perception of the PT4A intervention project? Probe:
  - What parts of the project did you like? Why?
  - What part of the project didn't you like? Why?
  - Parts of the project that were easily carried? What made it easy?
  - Parts of the project that were difficult to carry out? What made it difficult?
- 3. Now I would like you to share your experiences of the difference components of the PT4A intervention. How was your experience of;
  - Delivering HTN medication to individuals living with HTN?

- Providing psychological support to individuals living with hypertension at the community level
- Recording health information of the individuals receiving hypertension medication at the community on the mobile device (Probe: quality of care, provider-patient communication, privacy and confidentiality)
- Facilitating the doctor and the patient to have a clinical meeting using a mobile device at the community level (Probe: quality of care, provider-patient communication, privacy and confidentiality)
- 4. In what ways did the PT4A intervention affect the management of hypertension in the community?

#### Probe:

- How did it affect medication adherence for individuals living with hypertension?
- How did it affect clinic adherence for individuals living with hypertension?

### E. Mobile device.

Now let us talk more about the mobile device you used to deliver these health services to individuals living with hypertension at the community.

5. What was your perception about the mobile device you used as you delivered the PT4A intervention in the community

#### Probe:

- What did you like about the mobile device?
- What didn't you like about the mobile device?
- 6. What mobile device features were useful in implementing the PT4A intervention?

#### Probe:

- Content
- Data flow
- Connectivity
- 7. What mobile device features were not useful in implementing the PT4A intervention? Probe:
  - Content
  - Data flow
  - Connectivity
- 8. What was your perception about the mobile payment mode used to pay for the hypertension medications in the PT4A intervention?

#### Probe:

- What did you like about the mobile payment?
- What didn't you like about the mobile payment?
- 9. How did the use of a mobile device impact the delivery of hypertension services at the community?

PT4A Protocol 1.4 7<sup>th</sup> November, 2022

### F. Peers.

Following your experience as a peer in the PT4A project, I would now like us to talk about the qualities of a peer who would lead the delivery of PT4A intervention at the community.

10. What characteristics would be important for a peer to have if they were to lead the PT4A intervention in the community

#### Probe:

- Age
- Gender
- Personality
- Academic qualification
- Skill
- 11. What are your perceptions about the training you received from PT4A facilitators? Probe:
  - How relevant was the training in preparing you to conduct your duties as a peer in the PT4A intervention?
  - How adequate was the training in accomplishing your duties as a peer in the PT4A intervention?
  - What additional training aspects should be considered in the future for peers in the PT4A intervention?

# G. Recommendation for improving the PT4A project

We are about to end our discussion today. But before we end, we would like to hear about some of your recommendations for improving the proposed peer-led project to support individuals living with hypertension.

- 12. What is your perception about the uptake of this peer led project in your facility?
- 13. Would you recommend this peer-led project to other individuals living with HTN? Why
- 14. What would be your recommendation for improving this peer-led project? Probe:
  - Parts of the project that could be improved. How?
- 15. What would make this peer led project acceptable in the community?
- 16. What would make this peer-led project sustainable in the community?
- H. Closing

We have now come to the end of our discussions today. Thank you for your time and participation. We very much appreciate your comments, discussion, and input. We plan to take into account everything that was said today as we continue to improve the services we offer to your community.

Do you have any questions related to our discussion today?

## NB: Before ending

- Remind participants about the confidentiality of the interview.
- Ask if there is anything that wasn't raised that should have been that is important to know in understanding their perception about the peer-led intervention.

- Offer lunch stipend and provide contact information for any future questions they may have.
- Thank participants once again for their time.

Peers and Technology for Adherence, Access, Accountability, and Analytics (PT4A) Study Study Instrument: Focus Group Discussion (FGD) Guide for Design Team- Meeting 6.

| FGD moderator: | _ |
|-----------------|---|
| FGD note taker: | |
| Date://2022 | |
| County: | |
| Start Time: | |
| End Time: | |

#### FGD:

- Inform the participants about the study guided by the study information sheet.
- Provide participants with an opportunity to ask questions.
- Obtain written consent from each participant privately. (2 copies per participants)
- Provide each participant with a copy of their signed informed consent form.
- Complete the demographic survey for each participant privately.

# **Demographic Survey**

| Indicate or insert your responses as necessary | | | | |
|---|---|---|---|---|
| 1. Study ID: | | | | |
| 2. State your age (Years) | | | | |
| 3. Sex | Male | Female | | |
| 4. Where are you from? | Uasin-Gishu<br>County | Trans-Nzoia County | | Bungoma County |
| 5. Which group are you representing in the design team? | Health care<br>Team | Patients<br>Team | Peers<br>Team | Other (specify) |
| 6. How many design team meetings did you attend? | | | | |

NB: To be completed for each participant

# Focus Group Discussion Guide <u>Design Team</u>

**Opening Remarks:** Human-centered design is a creative approach to problem solving. It emphasizes issues that are important to community stakeholders rather than leadershipor administrators. This design process is focused on understanding the needs of the community, generating many ideas from different perspectives, building tangible prototypes, and iteratively improving the solution based on stakeholder feedback.

PT4A Protocol 1.4 7<sup>th</sup> November, 2022

During our Design Team meetings, we worked through phases of Inspiration, Brainstorming, Conceptualization, Creation, and Iteration. Through this process, we have learned much about the human-centered design methods and how they may be used tocreate a combined health information technology (HIT) and peer support program for PT4A. We have asked you to participate today because you have been a part of the PT4A Design Team. The purpose of this discussion is to reflect on your experience during the design process and provide feedback to the facilitators.

## **FGD** rules

Before we start, I would like as to you mention some of the rules that will guide our discussion

- 11. There are no right or wrong answers. We expect that you will have differing points of view. Please feel free to share your point of view even if it differs from what others have said.
- 12. We are recording this session as we discussed, because we do not want to miss any of your comments. No names will be included in any reports. Your comments are confidential. Please speak loudly for I want to be accurate in capturing what you say.
- 13. Don't feel like you have to respond all the time. But if you want to follow up on something that someone has said, you want to agree, or disagree, or give an example, feel free to do that.
- 14. I am here to ask questions, listen, and make sure everyone has a chance to share. We're interested in hearing from each of you. So if you are talking a lot, I may ask you to give others a chance. We just want to make sure all of you have a chance to share your ideas.
- 15. If you have a cell phone, please put it on quiet mode.

## A. DESIGN TEAM EXPERIENCE

- 1. Reflecting back to our first meeting, what is your understanding of human-centered design?
  - o Probe:
  - What were the goals of the design team?
- 2. Why did you volunteer to join the Design Team for PT4A?
  - o Probe:
  - What were your expectations for this design process?
  - Did this design process meet your expectations? Why or whynot?

PT4A Protocol 1.4 7<sup>th</sup> November, 2022

- 3. What have you learned during the human-centered design process?
  - o Probe:
  - What have you learned about yourself?
  - What have you learned about others in this group?
  - What have you learned about your community?
  - What have you learned about the health system?
- 4. Do you think that you will use what you have learned during the design process in the future? Please explain.
- 5. Often in group discussion, some participants may speak up and express opinions more than others. To what extent did every member of the DesignTeam participate equally in discussion?

#### o Probe:

- How have we succeeded to encourage participation from everyone in the group?
- What challenges have we faced in encouraging participation from everyone in the group?
- Were the opinions of each participant considered equally?Please explain.
- 6. Often in group discussion, there are times when there is disagreement between participants. How were disagreements addressed on the Design Team?

#### o Probe:

- When disagreements occurred, did the Design Team reach aconsensus before moving on? Please explain.
- 7. Reflecting on our work so far, to what extent did the Design Team incorporate:feedback from the community during the design process?
- 8. Reflecting on our work so far, to what extent did the Design Team incorporatefeedback from the PT4A investigators during the design process?
- 9. How do you feel about the current intervention model?

# Probe:

- How confident are you that it meets the original goals of ourdesign team?
- What are your thoughts about how this intervention was received by patients?
- What are your thoughts about how this intervention was received by providers and other health care workers?

# **B. RECOMMENDATION FOR IMPROVING HCD MEETINGS.**

10. What would be your recommendation for improving these design team meetings?

# C. CLOSING

Thank you for your time and participation. We very much appreciate your.Comments, discussion, and input. We plan to consider everything that was said today as we continue to improve the services we offer to your community.

Do you have any questions related to our discussion today?